#### Worldwide Clinical Trials Controlled Quality Management Document Sponsor: Xeris Pharmaceuticals Inc.

WORLDWIDE

**Protocol Number: DPI-201** 

## STATISTICAL ANALYSIS PLAN - TABLES, FIGURES AND LISTINGS SHELL **APPROVAL**

Study name: DPI-201: A Phase 2, Single-Dose, Randomized, Open-Label,

Active-Controlled. Crossover, Pharmacodynamic. Pharmacokinetic Comparative Study of a Novel Pramlintide-Insulin Co-Formulation in Adults with Type 1 Diabetes Mellitus

Statistical Analysis Plan (SAP)

Version being approved:

Version 1.0 / 14NOV2019

Tables, Figures and Listings

Table Shells version 1.0 / 14NOV2019 (TFL) Shell version being Figure Shells version 1.0 / 14NOV2019 approved: Listing Shells version 1.0 / 14NOV2019

The above SAP / TFL Shell has been reviewed and approved by Worldwide:

Name of Author:

**Tuomas Kemppainen** 

Position:

Senior Statistician / Biostatistics

Signature:

Tun Koo

Signer Name: Tuomas Kemppainen

DocuSigned by:

Signing Reason: I have reviewed this document Signing Time: 15-Nov-2019 | 09:21:11 GMT -Nov-2019 | 09:21:19 GMT -1555D305747C4F488CA546AD81C72A6E

Date:

Name of Reviewer:

Ioulietta Mulligan

DocuSigned by: Ioulietta Mulligan

Position:

**Manager / Biostatistics** 

Signature:

Signer Name: Ioulietta Mulligan

Signing Reason: I have reviewed this document Signing Time: 15-Nov-2019 | 13:58:23 GMT

Date:

15-Ney-79402D674683882746FE31684871

QMD Ref: Worldwide-TMP-ST-037-2.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

Confidentiality Statement



WORLDWIDE

Sponsor:

Xeris Pharmaceuticals Inc.

Protocol Number:

**DPI-201** 

## STATISTICAL ANALYSIS PLAN - TABLES, FIGURES AND LISTINGS SHELL APPROVAL

The above SAP / TFL Shell has been reviewed and approved by the Sponsor:

Name of Sponsor Medical:

Khaled Junaidi

Position:

**Medical Director** 

Signature:

Date:

14 Nov 2019

Name of Sponsor Clinical:

Joy Geallis on behalf of David Sequeira

Position:

Senior Manager, Clinical Operations

Signature:

Date:

14-NOV-2019

QMD Ref: Worldwide-TMP-ST-037-2,0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001



Sponsor:

Xeris Pharmaceuticals Inc.

Protocol Number:

DPI-201

## STATISTICAL ANALYSIS PLAN - TABLES, FIGURES AND LISTINGS SHELL APPROVAL

The above SAP / TFL Shell has been reviewed and approved by the Sponsor:

Name of Sponsor

Aziz Alam

Regulatory:

Position:

Senior Director, Regulatory Affairs

Signature:

Date:

4 NOV 2019

Name of Sponsor

**Nicole Close** 

Statistician:

Position:

**Head of Biometrics** 

Signature:

Data:

QMD Ref: Worldwide-TMP-ST-037-2.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

# WORLDWIDE Sponsor: Xeris Pharmaceuticals, Inc. Protocol Number: DPI-201 STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

## Statistical Analysis Plan

Title: Phase 2, Single-Dose, Randomized, Open-Label, Active-Controlled, Crossover, Pharmacodynamic, and Pharmacokinetic Comparative Study of a Novel Pramlintide-Insulin Co-Formulation in Adults with Type 1 Diabetes Mellitus

Protocol Number: DPI-201

Protocol Version: 3.0 / 06SEP2019

SAP Version 1.0

SAP Issue Date: 14-NOV-2019

SAP Author: Tuomas Kemppainen, MSc

**Previous SAP Versions** 

No previous versions

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

# Worldwide Clinical Trials Controlled Quality Management Document Sponsor: Xeris Pharmaceuticals, Inc. Protocol Number: DPI-201 STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

## **SAP Amendments Before Database Lock**

| Version | Issue Date | Section | Revision / Addition | Rationale |
|---|---|---|---|---|
| 0.1 | 28-AUG-2019 | | | First draft for internal |
| | | | | review. |
| 0.2 | 02-SEP-2019 | | | First draft for Sponsor |
| | | | | review. |
| 0.3 | 19-SEP-2019 | | | Second draft for Sponsor |
| | | | | review. Including TFL |
| | | | | shells. |
| 0.4 | 08-OCT-2019 | | | Pre-final version. |
| 1.0 | 08-NOV-2019 | | | Version 1.0 |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

#### **Confidentiality Statement**



Sponsor: Xeris Pharmaceuticals, Inc.
Protocol Number: DPI-201

#### STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

## **Table of Contents**

| 1 | INI | RODUCTION | / |
|---|---|---|---|
| 2 | STU | DY OBJECTIVES | 7 |
| | 2.1 | Primary Objective | 7 |
| | | Secondary Objectives. | |
| 3 | | POINTS | |
| | | Primary Endpoint | |
| | | Secondary Endpoints | |
| | 3.2.1 | Safety Endpoints | |
| | 3.2.2 | | |
| 4 | SAN | MPLE SIZE | |
| 5 | | NDOMIZATION | |
| 6 | PLA | NNED ANALYSES1 | 0 |
| | 6.1 | Analysis Sets | 0 |
| | 6.1.1 | Enrolled Set | |
| | 6.1.2 | Randomized Set1 | 0 |
| | 6.1.3 | Safety Analysis Set | 0 |
| | 6.1.4 | PD Analysis Set | 0 |
| | 6.2 | Derived Data | 0 |
| | 6.2.1 | Age | 0 |
| | 6.2.2 | Race1 | 1 |
| | 6.2.3 | Baseline | 1 |
| | 6.2.4 | Duration / Study Day / Time | 1 |
| | 6.2.5 | Conventions for Missing and Partial Dates | 1 |
| | 6.2.6 | Missing / Partial Start / Stop Date of Adverse Events (AE) and Concomitant | |
| | Medi | cations1 | 1 |
| | 6.2.7 | $\mathcal{E}$ | |
| | 6.2.8 | Missing Diagnosis Dates | 3 |
| | 6.2.9 | Exposure to Study Drug | 3 |
| | 6.2.1 | | |
| | 6.2.1 | J 1 | |
| | 6.2.12 | | |
| | 6.3 | Conventions | 5 |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

#### **Confidentiality Statement**



Sponsor: Xeris Pharmaceuticals, Inc.

Protocol Number: DPI-201

## STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| | 6.3.1 | Decimal Places | 16 |
|----|---------|--------------------------------------|-----|
| 6. | 4 Su | bject Disposition | 16 |
| 6. | 5 Pr | otocol Deviations | 17 |
| 6. | 6 Ba | aseline Comparability | 17 |
| 6. | 7 M | edical History | 17 |
| 6. | 8 Pr | ior/Concomitant Medications | 18 |
| 6. | 9 Ex | xposure to Study Drug | 18 |
| 6. | 10 Tı | reatment Compliance | 18 |
| 6. | 11 Ef | ficacy Analyses | 18 |
| | 6.11.1 | Primary Endpoint | 18 |
| | 6.11.2 | Multiplicity | 19 |
| 6. | 12 Pł | narmacodynamic Analyses | 19 |
| 6. | 13 Sa | ıfety Analyses | 19 |
| | 6.13.1 | Adverse Events | 19 |
| | 6.13.2 | Laboratory Data | 20 |
| | 6.13.3 | C-Peptide and HbA1c | 20 |
| | 6.13.4 | Urine Drug Screen | 21 |
| | 6.13.5 | Urine Pregnancy Test | 21 |
| | 6.13.6 | Vital Signs | 21 |
| | 6.13.7 | Electrocardiogram Data | 21 |
| | 6.13.8 | Physical Examination. | 22 |
| | 6.13.9 | Draize Scale | 22 |
| | 6.13.10 | Injection Site Discomfort Assessment | 22 |
| | 6.13.11 | Hypoglycemic Events | 23 |
| 7 | INTE | RIM ANALYSIS | 25 |
| 3 | DATA | SAFETY MONITORING BOARD ANALYSIS | 25 |
| ) | CHAN | IGES TO PLANNED PROTOCOL ANALYSIS | 25 |
| 0 | REFE | RENCES | 26 |
| | | OF TABLES FIGURES AND LISTINGS | 2.7 |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

**Confidentiality Statement** 

## WORLDWIDE Sponsor: Xeris Pharmaceuticals, Inc. Protocol Number: DPI-201

STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

#### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|---|---|
| AE | adverse event |
| AESI | adverse event of special interest |
| ALT | alanine aminotransferase |
| ANOVA | analysis of variance |
| AOC | area over the curve |
| AST | aspartate aminotransferase |
| AUC | area under the concentration-time curve |
| AUC <sub>0-90</sub> | area under the concentration-time curve from 0 to 90 minutes post-dosing |
| AUC <sub>0-180</sub> | area under the concentration-time curve from 0 to 180 minutes post-dosing |
| AUC <sub>0-360</sub> | area under the concentration-time curve from 0 to 360 minutes post-dosing |
| BGM | blood glucose measurement |
| BMI | body mass index |
| BP | blood pressure |
| CLIA | Clinical Laboratory Improvement Act |
| C <sub>max</sub> | maximum plasma concentration |
| CRF | case report form |
| CRO | contract research organization |
| eCRF | electronic case report form |
| ECG | electrocardiogram |
| EDC | electronic data capture |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practices |
| GLP-1 | Glucagon-like peptide-1 |
| HbA1c | glycated hemoglobin |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| HR | heart rate |

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |



Sponsor: Xeris Pharmaceuticals, Inc.

Protocol Number: DPI-201

## STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| Abbreviation | Definition |
|---|---|
| IB | Investigator's Brochure |
| I:C | insulin-to-carbohydrate |
| ICF | informed consent form |
| IEC | Independent Ethics Committee |
| ICH | International Conference on Harmonisation |
| IME | important medical event |
| IND | Investigational New Drug |
| IRB | institutional review board |
| IUD | intra-uterine device |
| IWRS | Interactive Web Response System |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NRS | Numeric Rating Scale |
| PD | pharmacodynamics(s) |
| PE | physical examination |
| PK | pharmacokinetic(s) |
| PT | Preferred Term |
| PRAM9 | Co-formulation of a fixed-ratio combination of 9 µg pramlintide per unit of regular insulin |
| RBC | red blood cells |
| SAE | serious adverse event |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| SD | standard deviation |
| SE | standard error |
| SOC | System Organ Class |
| T1D | Type 1 diabetes mellitus |
| TEAE | treatment-emergent adverse event |
| T <sub>max</sub> | time to maximum plasma concentration |
| ULN | upper limit of normal |
| WHO | World Health Organization |

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
|---|---|

**Confidentiality Statement** 

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| CLINICAL TRIALS | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

#### 1 INTRODUCTION

This document details the planned statistical analyses for the Xeris Pharmaceuticals, Inc., protocol "DPI-201" study titled "A Phase 2, Single-Dose, Randomized, Open-Label, Active-Controlled, Crossover, Pharmacodynamic, and Pharmacokinetic Comparative Study of a Novel Pramlintide-Insulin Co-Formulation in Adults with Type 1 Diabetes Mellitus".

The proposed analyses are based on the contents of the final version 3.0 of the protocol (dated 06-SEP-2019).

Analyses for pharmacokinetic (PK) parameters will be covered in a separate Statistical Analysis Plan (SAP).

This is a randomized, open-label, active-controlled, single-dose, 3-treatment, 3-period, 3-way crossover, comparative PD, and PK inpatient study in adults with Type 1 Diabetes Mellitus (T1D).

Most people with diabetes are still unable to achieve glycemic targets with sole insulin therapy alone, particularly after mealtime. Physiologic restoration of the hormonal responses during meals, via pramlintide and insulin, has been demonstrated to reduce postprandial hyperglycemia and to improve blood glucose time in range.

The synergy between insulin and pramlintide provides improved glucose control while reducing meal-time insulin requirements. Reduced insulin utilization may also reduce the effects associated with long-term insulin use such as weight gain and higher risks of hypoglycemia.

A pramlintide-insulin co-formulation may help reduce the burden associated with co-administration (e.g., reduce the number of injections per day). Additionally, coformulations of pramlintide and insulin may also improve treatment compliance and persistency.

#### 2 STUDY OBJECTIVES

## 2.1 Primary Objective

The primary objective of this study is to evaluate the PD properties of a single dose of PRAM9 (referred to as XP-3924 in tables, listings, figures) compared to single doses of regular insulin and regular insulin plus pramlintide (co-administered as separate injections) in adults with T1D.

## 2.2 Secondary Objectives

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without | |
| prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures | |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE | Sponsor: | Xeris Pharmaceuticals, Inc. |
| CLINICAL TRIALS | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

The secondary objectives of this study are to evaluate the safety and PK profiles of a single dose of PRAM9 compared to single doses of regular insulin and regular insulin plus pramlintide (coadministered as separate injections) in adults with T1D.

#### 3 ENDPOINTS

## 3.1 Primary Endpoint

Analysis of the primary endpoint will be performed using the PD Analysis Set. The PD effects upon plasma glucose levels will be compared between the treatments as defined by the following primary endpoint:

• Area under the curve area from administration to 180 min (AUC<sub>0-180</sub>) (mg/dL × minutes) for plasma glucose > 180 mg/dL.

## 3.2 Secondary Endpoints

## 3.2.1 Safety Endpoints

All safety analyses will be performed using the Safety Analysis Set.

The following safety variables will be compared between the treatments:

- Incidence of adverse events (AEs) and serious adverse events (SAEs)
- Change from baseline in laboratory safety variables
- Change from baseline in vital sign measurements
- Change from baseline in body weight
- Local tolerability assessments, including:
  - Incidence of erythema and or edema formation at site of injection assessed using the Draize scale (See Protocol Appendix 1)
  - Subjective injection site discomfort as reported by subjects using a 11-point Numeric Rating Scale (NRS) (See Protocol Appendix 2).
- Hypoglycemic events
  - o Time to IV Dextrose administration from study drug administration
  - o Time to hypoglycemic event from study drug administration
  - o Time to resolution of hypoglycemic event from IV Dextrose administration
  - o Proportion of subjects reaching euglycemia after IV Dextrose administration
  - Average amount of IV Dextrose

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without | |
| prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. | |

## WORLDWIDE SPONSOR: DPI-201 STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

## 3.2.2 Pharmacodynamic Endpoints

All PD analyses will be performed using the PD Analysis Set. The following variables will be compared between the treatments:

- Mean proportional time with plasma glucose X mg/dL (during 0-t minutes post-injection of study drug), where X=(<54, <70, >180, >250) and t=(90, 180, 360) leading to 12 parameters. The primary PD endpoint will be X='>180' and t='180'.
- Mean proportional time after glucose challenge for plasma glucose levels between 126 to 180 mg/dL (during 40 to 180 minutes post-injection of study drug)
- AUC<sub>0-t</sub> (mg/dL × minutes) for plasma glucose X mg/dL, where X=(>180, >250) and t=(90, 180, 360) leading to 6 parameters.
- AOC<sub>0-t</sub> (mg/dL × minutes) for plasma glucose X mg/dL, where X=(<54, <70) and t=(90, 180, 360) leading to 6 parameters.
- Plasma glucose C<sub>max</sub> and T<sub>max</sub>.

#### 4 SAMPLE SIZE

Up to 21 subjects will be qualified for the study and will complete the overnight stay as part of Visit 2 to ensure that 18 total subjects are randomized to a study treatment sequence. The target of 18 randomized subjects is considered sufficient to allow an initial evaluation of PK/PD response and safety of the novel pramlintide-insulin formulation. Formal sample size calculations were not conducted.

#### 5 RANDOMIZATION

On the morning of Visit 2, subjects will be randomized into the appropriate treatment sequence order to receive each of the 3 study treatments (PRAM9, regular insulin, and co-administered regular insulin plus pramlintide). The study statistician will create the randomization sequence using random permuted block methodology. Study drug administration randomization sequences are as follows:

| Cohort | Period 1 | Period 2 | Period 3 |
|---|---|---|---|
| 1 | PRAM9 | Regular insulin | Regular insulin + pramlintide |
| 2 | Regular insulin | Regular insulin + pramlintide | PRAM9 |
| 3 | Regular insulin + pramlintide | PRAM9 | Regular insulin |
| 4 | PRAM9 | Regular insulin + pramlintide | Regular insulin |
| 5 | Regular insulin | PRAM9 | Regular insulin + pramlintide |
| 6 | Regular insulin + pramlintide | Regular insulin | PRAM9 |

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |
| TI: 1 4: 4 CW 11:1 CI: 1T:1 I 4 1 1:4 1 1:4 1 1:4 1 | |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

#### 6 PLANNED ANALYSES

No statistical analysis plan (SAP) prepared in advance of the data can be absolutely definitive and the final Clinical Study Report (CSR) may contain additional tables or statistical tests if warranted by the data obtained. The justification for any such additional analyses, or deviations from this SAP, will be fully documented in the final clinical study report (CSR).

## 6.1 Analysis Sets

Subjects excluded from the analysis sets and the reason for their exclusion will be listed in Appendix 16.2 of the CSR.

Analyses performed on the Safety Analysis Set will use the actual treatment received. All other populations will use the randomized treatment.

#### 6.1.1 Enrolled Set

The Enrolled Set includes all subjects who gave informed consent.

#### 6.1.2 Randomized Set

The Randomized Set includes all subjects who were randomized to the treatment sequence.

## 6.1.3 Safety Analysis Set

The Safety Analysis Set includes all randomized subjects who received any study drug.

## 6.1.4 PD Analysis Set

The PD Analysis Set includes all subjects from Safety Analysis Set who had blood glucose measured at pre-dose and 180 minutes post-dose, and at least one time point between pre-dose and 180 minutes post-dose.

#### **6.2** Derived Data

This section describes the derivations required for statistical analysis. Unless otherwise stated, variables derived in the source data will not be re-calculated.

## **6.2.1** Age

Age at screening will be collected in the CRF.

| Governing QMD: Worldwide-SOP-ST-001 |
|---|
| Confidentiality Statement |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. |
| ı |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE<br>CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

## 6.2.2 Race

Where more than one race category has been selected for a subject, these race categories will be combined into a single category labeled "Multiple Race" in the summary tables. The listings will reflect the original selected categories.

#### 6.2.3 Baseline

The baseline is defined as the last non-missing value (either scheduled, unscheduled or repeat) that is collected before dosing of each treatment period.

## **6.2.4 Duration / Study Day / Time**

Study day will be calculated as the number of days from first dose of the study drug on period 1 (Study Day 1).

- date of event date of first dose of study drug on period 1 (+ 1), for events on or after first dose
- date of event date of first dose of study drug on period 1, for events before first dose.

## 6.2.5 Conventions for Missing and Partial Dates

All rules explained below for partial / missing dates will be followed unless contradicted by any other data recorded on the electronic Case Report Form (eCRF).

All dates presented in the individual subject listings will be as recorded on the eCRF (i.e., not completed as per the below rules).

## 6.2.6 Missing / Partial Start / Stop Date of Adverse Events (AE) and Concomitant Medications

Missing and partial start and stop date will be imputed for analysis purposes as follows.

#### Partial or missing stop date will be imputed as follows:

If the stop date is completely missing and the event has resolved, or the subject has stopped taking the concomitant medication, the stop date will be imputed as the date of the subject's last clinic visit in the study.

• If only the year is known, the stop date will be imputed as "31-Dec" of that year or as the date of the subject's last clinic visit in the study if in the same year.

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. | |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE<br>CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

• If the month and year are known, the stop date will be imputed as the last day of that month unless the stop date corresponds to the same month as the subject's last clinic visit in which case the date of subject's last clinic visit in the study will be used instead.

#### Missing start date will be imputed as follows:

- If the stop date occurs on or after the start of study drug or the event / concomitant medication is ongoing, the start date will be imputed as the date of the first dose of study drug.
- If the stop date occurs before the start of study drug, the start date of the event / concomitant medication will be imputed as the subject's screening date or the stop date of the event / concomitant medication whichever is earlier.

## Partial start date (year present, but month and day missing)

- If the stop date occurs on or after the start of study drug or the event / concomitant medication is ongoing, and the year is the same as the year of first dosing the start date will be imputed as "01-Jan" of the same year or the date of the first dose of study drug whichever is latest. If the year is different from the year of first dosing "01-Jan" will be used.
- If the stop date occurs before the start of study drug, the start date of the event / concomitant medication will be imputed as the "01-Jan" of the same year.

#### Partial start date (month and year present, but day missing)

- If the stop date occurs on or after the start of study drug or the event / concomitant medication is ongoing, the start date will be imputed as the first day of the same month and year unless this partial start date is in same month as the first dose of study drug in which case the date of first dose of study drug will be used.
- If the stop date occurs before the start of study drug, the start date will be imputed as the first day of the month and year of the partial stop date.

If the start time is missing it will be imputed only in the case where the start date of the concomitant medication / event corresponds to the date of the study drug dosing. The time will be imputed as the same time as the study drug dosing for each period. In all other cases the time will not be imputed.

## **6.2.7** Missing Last Dates of Study Drug Dosing

Study drug dosing dates and times will not be imputed. This is single dose cross-over study and the dosing information need to be collected in the CRF.

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without | |
| prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. | |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

## **6.2.8** Missing Diagnosis Dates

If the month and year are present but the day is missing, the diagnosis date will be set to first day of the relevant month. If only the year is recorded the diagnosis date will be set as "01-Jan" for that year.

## 6.2.9 Exposure to Study Drug

Exposure to study drug will not be calculated as this is a single dose study.

#### **6.2.10** Inexact Values

In the case where a laboratory or PD variable is recorded as "> x", " $\geq$  x", " $\leq$  x" or " $\leq$  x", a value of x will be taken for analysis purposes.

## 6.2.11 Primary Endpoint and PD Parameters

The figure below is presented only to show the idea of the calculation of PD parameters and the shape of the curve is based on dummy data. PD parameters will be calculated using linear trapezoidal rule.

WORLDWIDE CLINICAL TRIALS Sponsor: Xeris Pharmaceuticals, Inc.
Protocol Number: DPI-201

STATISTICAL ANALYSIS PLAN. PHASE 2-3-4



#### $AUC_{0-t}$ (mg/dL × minutes) for plasma glucose > XXX mg/dL

From the above example figure the area under the curve (AUC) for concentration > 5 is calculated as follows:

$$(60-37.5)(0+3)/2 + (120-60)(3+5)/2 + (180-120)(5+3)/2 + (240-180)(3+0)/2 = 33.75 + 240 + 240 + 90 = 603.75$$

#### Mean proportional time for plasma glucose < XXX mg/dL

From the above example figure the mean proportional time for concentration < 5 is calculated as follows:

$$(37.5 - 0 + 360 - 240) / (360-0) = 157.5 / 360 = 43.75\%$$

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without | |
| prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. | |

REF: Worldwide-TMP-QA-001f-1.3

# WORLDWIDE STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

## AOC<sub>0-t</sub> (mg/dL × minutes) for plasma glucose < XXX mg/dL

From the above example figure the area over the curve (AOC) for concentration < 5 is calculated as follows:

$$(37.5-0)(5+0)/2 + (300-240)(0+3)/2 + (360-300)(3+4) = 93.75 + 90 + 210 = 393.75$$

#### **6.2.12** Unscheduled Visits

Only scheduled post-baseline values will be tabulated. Post-baseline repeat / unscheduled assessments will not be tabulated, although these post-baseline assessments will be listed in the relevant appendices to the CSR.

#### 6.3 Conventions

All data listings, summaries, figures and statistical analyses will be generated using SAS version 9.4 or higher<sup>1</sup>.

Summaries will be presented by treatment group or treatment sequence as appropriate. Treatment group labels will be displayed as follows:

- XP-3924
- Regular Insulin
- Regular Insulin + Pramlintide
- Overall

Treatment sequence labels will be displayed as follows:

- A-B-C
- B-C-A
- C-A-B
- A-C-B
- B-A-C
- C-B-A
- Overall

Where

A = XP-3924

B = Regular Insulin

C = Regular Insulin + Pramlintide.

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-S |
|---|
|---|

#### **Confidentiality Statement**

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE<br>CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

Listings will be sorted in the following order treatment group / sequence, subject, parameter, and visit unless otherwise stated. All data will be listed, subjects who were not randomized will be displayed after the randomized treatment / sequence groups.

Continuous variables will be summarized by the number of non-missing observations, mean, median, standard deviation, and minimum and maximum. For all tabulations of changes from baseline data, the lower and upper 95% confidence limits for the mean for the individual treatments will be given. Summaries for PD parameters will also include 95% confidence interval, coefficient of variation (%CV) and quartiles (Q1 and Q3).

Categorical variables will be summarized by presenting the frequency and percent. Percentages will be based on the number of non-missing observations or the subject population unless otherwise specified. For each variable, all categories will be shown. Zero frequencies (but not the percent) within a category will be presented.

#### **6.3.1** Decimal Places

Decimal places for derived data described in section 6.2 will be determined by the scale of measurement unless otherwise stated. No decimal places will be displayed if the smallest calculated value is  $\geq 100$ ; 1 decimal place will be displayed when the smallest value is within the interval (10, 100), with 10 being inclusive; 2 decimal places will be displayed when the smallest value is within (1, 10), with 1 being inclusive; and so on for even smaller scales of measurement.

Derived data where it is known in advance the result will be an integer for example day, month, year, number of days and total scores (for rating scales) will be presented with zero decimal places.

Means, medians and percentiles will be displayed to one more decimal place than the data, dispersion statistics (e.g. standard deviation) will have two more decimal places, and the minimum and maximum will be displayed to the same number of decimal places as reported in the raw data. Percentages will be displayed with one decimal place.

P-values will be quoted to 3 decimal places. P-values < 0.001 will be presented as p<0.001. Where this value is less than 0.05, 0.01 or 0.001, attention will be drawn to this fact using the conventional "\*", "\*\*" or "\*\*\*" annotation, respectively.

## 6.4 Subject Disposition

Subject disposition will be summarized as follows:

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
| Confidentiality Statement | |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without | |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

- The number of subjects who failed screening and the reasons for failure will be tabulated for enrolled set.
- The number of subjects included in the analysis sets will be summarized by treatment sequence and overall for the enrolled set.
- The number of early withdrawals and the reasons for withdrawals will be tabulated by treatment sequence and overall for the enrolled set.

#### **6.5** Protocol Deviations

Protocol Deviations will be summarized in frequency table by treatment sequence (including overall).

A listing of protocol deviations will be provided within Appendix 16.2 of the CSR.

## **6.6** Baseline Comparability

The comparability of treatment sequences with respect to subject demographics and baseline characteristics will be assessed in a descriptive manner, but no formal statistical testing will be performed.

Standard continuous or categorical variable summaries will be presented by randomized treatment sequence and overall for the following variables based on the Safety Analysis Set.

- Demographic data
  - o Age
  - o Sex (Male, Female)
  - o Childbearing potential for Female (Yes, No)
  - Race (White, Black or African American, Asian, American Indian or Alaskan Native, Native Hawaiian or Other Pacific Islander)
  - o Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
  - o Height (cm)
  - Weight (kg)
  - $\circ$  BMI (kg/m<sup>2</sup>).

## 6.7 Medical History

Medical history will be coded using the Medical Dictionary of Regulated Activities (MedDRA) (version 22.0). All medical history will be presented by treatment sequence and overall for the Safety Analysis Set by primary system organ class and preferred term.

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-ST |
|---|
| Confidentiality Statement |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without |
| prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE<br>CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

## 6.8 Prior/Concomitant Medications

All prior/concomitant medications will be presented by treatment sequence and overall for the Safety Analysis Set. Prior medications are defined as all medications ending before the date of first dose of study drug. Concomitant medications are defined as medications taken on or after the date of first dose of study drug. Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary (version WHODrug Global B3 Mar 2019) and summarized using Anatomic Therapeutic Chemical (ATC) Level 4 and preferred term.

## 6.9 Exposure to Study Drug

Study drug administration will be summarized in frequency table by treatment sequence, treatment period and treatment group for the Safety Analysis Set.

## 6.10 Treatment Compliance

Not applicable.

## 6.11 Efficacy Analyses

All statistical tests will be performed using a two-tailed 5% overall significance level, unless otherwise stated. All comparisons between treatments will be reported with 95% confidence intervals for the difference.

## 6.11.1 Primary Endpoint

 $AUC_{0-180}$  (mg/dL × minutes) for plasma glucose > 180 mg/dL will be summarized using descriptive statistics by period (including overall) and treatment group in PD Analysis Set.

Treatment groups will be compared using analysis of variance (ANOVA) model including sequence, period and treatment as fixed effects and subject within sequence as random effect. The hypothesis to be tested is as follows:

H<sub>0</sub>: Means are equal between treatment groups.

H<sub>a</sub>: Means are not equal across the treatment groups.

The SAS code for analysis is as follows:

```
proc mixed data=dataset order=internal;
class subject sequence period treatment;
model response=sequence period treatment / ddfm=kr;
random subject(sequence);
```

| 1 | OMD B C W. 11 '1 TM D CT 007 7 0 FCC ' 124 2010 | C ' OMD W II 'I COD CT ON |
|---|---|---|
| | QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
| | Confidentiality | Statement |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

```
lsmeans treatment / diff cl e;
ods output tests3=test1 lsmeans=lsm1 diffs=dif1;
run;
```

## 6.11.2 Multiplicity

All secondary endpoints and the supportive analyses will be considered as descriptive evidence of efficacy and will be analyzed without any procedures to account for multiple comparisons.

## **6.12 Pharmacodynamic Analyses**

The endpoints specified in section 3.2.2 (except plasma glucose  $T_{max}$ ) will be analyzed similarly to the primary endpoint in PD Analysis Set.

Plasma glucose  $T_{max}$  will be compared between treatment groups using Wilcoxon Signed Rank test. Comparison will be done separately for each pairwise comparisons between the treatment groups (PRAM9 vs. Regular Insulin, PRAM9 vs. Regular Insulin + Pramlintide, Regular Insulin vs. Regular Insulin + Pramlintide). The SAS code for analysis is as follows:

```
proc univariate data=paired1 mu0=0;
var diff;
run;
```

Where diff is the difference between the two compared treatment groups for each subject.

## **6.13 Safety Analyses**

The safety analyses will be presented by the treatment received for the Safety Analysis Set if not otherwise stated.

#### 6.13.1 Adverse Events

A treatment emergent adverse event (TEAE) is defined as:

- Any AE that has an onset on or after the first dose of study drug
- Any pre-existing AE that has worsened in severity on or after the first dose of study drug. The following rules will be used to assign a TEAE to a treatment group:
  - A TEAE will be assigned to the treatment received immediately before onset.
  - Any TEAE reported within the washout period between doses will be attributed to the previous treatment.
  - If the severity of a TEAE increases in a later period, the TEAE at the increased severity will be assigned to the treatment received immediately before the increase in severity.

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-ST-00 |
|---|
| Confidentiality Statement |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. |

REF: Worldwide-TMP-QA-001f-1.3

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

A treatment-related AE is defined as an AE as having suspected relationship to the study drug. If an AE has missing relationship it is assumed to be related to the study drug for analysis purposes.

Maximum severity (severe) will be assumed for an AE with missing severity.

Adverse Events will be coded using the Medical Dictionary of Regulated Activities (MedDRA) (version 22.0) primary system organ class and preferred term.

The following tables will be presented for AEs by treatment group and overall. Additionally, tables will be presented by treatment period and overall.

- Overall incidence and the number of:
  - o Any AEs
  - o TEAEs
  - o Treatment-Related TEAEs
  - Severe or life-threatening TEAEs
  - Serious TEAEs
  - o Treatment-Related Serious TEAEs
  - o SAEs leading to death
  - o TEAEs leading to early withdrawal.
  - o Serious TEAEs leading to early withdrawal.
- For the above AE categories tables including incidence and number of events will be presented by system organ class and preferred term.

All AEs will be listed.

## 6.13.2 Laboratory Data

Descriptive statistics of the observed values and change from baseline (continuous data) will be presented overall by visit for each hematology and serum chemistry parameter. Each measurement (continuous data) will be classed as below, within, or above normal range, based on ranges supplied by the laboratory used (Altasciences for PK and Worldwide for routine safety labs). Shift tables in relation to the normal range from baseline to each follow-up visit will be presented.

## 6.13.3 C-Peptide and HbA1c

C-Peptide and HbA1c will be collected only at screening visit.

Descriptive statistics of the observed values will be presented overall.

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-ST-00 |
|---|
| Confidentiality Statement |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. |

# WORLDWIDE STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 Worldwide Clinical Trials Controlled Quality Management Document Sponsor: Xeris Pharmaceuticals, Inc. Protocol Number: DPI-201

## 6.13.4 Urine Drug Screen

Urine drug screen will be collected only at screening visit and will include the following analytes: cocaine, THC, opiates, amphetamines, methamphetamine and phencyclidine.

Urine drug screen data will be listed only.

## **6.13.5** Urine Pregnancy Test

Urine pregnancy test data will be listed only.

## 6.13.6 Vital Signs

Descriptive statistics for observed values and changes from baseline in the following vital signs will be presented by treatment group (including overall) and visit:

- Systolic blood pressure (mmHg)
- Diastolic blood pressure (mmHg)
- Heart rate (bpm)
- Respiration rate (breath / min)
- Body temperature (degrees Celsius)
- Body weight (kg).

## 6.13.7 Electrocardiogram Data

ECG will be collected only at screening visit.

Descriptive statistics for observed values in the following ECG variables will be tabulated overall at screening:

- PR Duration (ms)
- RR Interval (ms)
- QRS Duration (ms)
- QT Interval (ms)
- QTc Interval (ms)
- QTcF Interval (ms)
- QTcB Interval (ms)
- Ventricular Rate (bpm).

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|

#### **Confidentiality Statement**

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

Overall interpretation (Normal, Abnormal NCS, and Abnormal CS) will be presented overall at screening in frequency table.

## 6.13.8 Physical Examination

The body systems within the physical examination data at the end of the study will be summarized overall for the shift from baseline to the end of the study (Normal, Abnormal (NCS), Abnormal (CS), Not Done).

All physical examination data will be listed.

#### 6.13.9 Draize Scale

Draize scale will be presented by treatment group and overall by time point (30 min, 90 min and 360 min post-dose) in frequency table.

Data will be summarized for Erythema Formation:

- 0 No erythema
- 1 Very slight erythema
- 2 Well defined erythema
- 3 Moderate erythema
- 4 Severe erythema

#### and Edema Formation:

- 0 No edema
- 1 Very slight edema
- 2 Slight edema
- 3 Moderate edema
- 4 Severe edema

## **6.13.10** Injection Site Discomfort Assessment

Injection Site Discomfort Assessment includes:

- Numeric Rating Scale (NRS) for Injection Site Discomfort
  - o 11-point scale from 0 to 10
- 1a. How would you describe any discomfort you felt from the study drug? (Check all that apply):

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-ST-00 |
|---|
| Confidentiality Statement |
| This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures. |

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN, PHASE 2-3-4 | | |

- o None (Please ignore question 1b.)
- o Pain (eg, throbbing, soreness, muscle ache)
- Itching
- o Tingling, twitching, or numbness
- o Irritation (eg, burning, stinging)
- o Other
- 1b. About how long did the discomfort last after the injection? (Check one):
  - o Less than 1 minute
  - o 1-2 minutes
  - o 3-5 minutes
  - o 6-9 minutes
  - o at least 10 minutes (Please complete question 1c before leaving the clinic.)
- 1c. In total, how long did the discomfort last after the injection? (Please enter a number below):
  - o \_\_\_\_ Minutes

For NRS, descriptive statistics for observed values will be presented by treatment group (including overall) and time point (10 min, 30 min post-dose).

Questions 1a, 1b and 1c are answered only once after each dosing and will be presented in frequency tables (1a and 1b) and using descriptive statistics (1c) by treatment group (including overall).

## 6.13.11 Hypoglycemic Events

Time to event endpoints will be analyzed by comparing the survivor functions between treatment arms using Kaplan-Meier methodology. Estimates and 95% confidence intervals for the median time to event, and 25th and 75th percentiles will be reported. Log-rank test will be performed to test the homogeneity of survival curves between the treatment groups.

Kaplan-Meier plots by treatment group will be provided including the number of subjects remaining at risk at each time point.

The SAS code for analysis is as follows:

```
proc lifetest data=dataset method=km outsurv=surv
plots=survival(atrisk=(0 to 50 by 5) /*cb=hw test*/);
time time*cens(1);
strata treatment / order=internal;
run;
```

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-ST-001

Confidentiality Statement

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE<br>CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

Where time is the time to the event and cens(1) is the censoring variable with censored records defined in brackets.

#### Time to IV Dextrose administration from study drug administration

Calculated as time in minutes from study drug administration to administration of IV Dextrose. If subject is not receiving IV Dextrose then subject will be censored at the start of glucose challenge or 4 hours after the study drug administration whichever is the earliest.

## Time to hypoglycemic event from study drug administration

Calculated as time in minutes from study drug administration to the start of hypoglycemic event. If subject is not having hypoglycemic event then subject will be censored at the start of glucose challenge or the time of next study drug administration or the follow-up visit in case of last treatment period whichever is the earliest.

#### Time to resolution of hypoglycemic event from IV Dextrose administration

Will be calculated only for subjects who experience hypoglycemic event. Calculated as time in minutes from administration of IV Dextrose to the time of resolution of hypoglycemic event. Resolution is defined and blood glucose reading crossing the 70 mg/dL threshold. Resolution timepoint will be estimated using linear estimation. Censoring will not be done as hypoglycemic events should be resolved before subjects are discharged from the clinic.

#### Proportion of subjects reaching euglycemia after IV dextrose administration

Proportion of subjects reaching the euglycemia (blood glucose >= 70 mg/dL) at 10, 20, 30 minutes post-IV-Dextrose-administration will be summarized in frequency table by treatment group.

#### **Average Amount of IV Dextrose**

Amount of IV Dextrose administered after hypoglycemic event will be summarized using descriptive statistics by treatment group.

Treatment groups will be compared using paired t-test. Comparison will be done separately for each pairwise comparisons between the treatment groups (PRAM9 vs. Regular Insulin, PRAM9 vs. Regular Insulin + Pramlintide, Regular Insulin vs. Regular Insulin + Pramlintide). The SAS code for analysis is as follows:

```
proc ttest data=paired1;
paired result1*result2;
run;
```

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|

**Confidentiality Statement** 

# Worldwide Clinical Trials Controlled Quality Management Document Sponsor: Xeris Pharmaceuticals, Inc. Protocol Number: DPI-201 STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

Where result1 and result2 are the doses for treatment groups.

#### 7 INTERIM ANALYSIS

No interim analyses are planned.

#### 8 DATA SAFETY MONITORING BOARD ANALYSIS

No data safety monitoring board (DSMB) analyses are planned.

#### 9 CHANGES TO PLANNED PROTOCOL ANALYSIS

Several PD parameters were added for mean proportional time with different cutoffs for plasma glucose levels and timepoints leading to total of 12 parameters. Similar update was done for AUC0-t parameters also leading to total of 12 different parameters.

Analysis for hypoglycemic events (time to IV Dextrose administration, time to hypoglycemic event, time to resolution of hypoglycemic event, proportion of subjects reaching euglycemia and average amount of IV Dextrose) were added.

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

| Worldwide Clinical Trials Controlled Quality Management Document | | |
|---|---|---|
| WORLDWIDE CLINICAL TRIALS | Sponsor: | Xeris Pharmaceuticals, Inc. |
| CLINICAL TRIALS | Protocol Number: | DPI-201 |
| STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 | | |

## 10 REFERENCES

1. SAS Institute Inc., Cary, NC, 27513, USA

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

## WORLDWIDE SPONSOR: SPONSOR: DPI-201 STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

## 11 LIST OF TABLES, FIGURES AND LISTINGS

The following table includes details of the tables, figures and listings to be included within each section of the eCTD. The eCTD section is shown in bold. The following validation methods maybe used:

- Independent programming of numbers and manual review of format (IP)
- Independent programming by statistician of numbers and manual review of format (Stat IP)
- Manual review (MR)
- Code review (CR)

| Table<br>Number | Table Title | Validation<br>Method | Shell<br>Number<br>(if repeat) |
|---|---|---|---|
| Items in bold | l are not table titles but references to the section headings v | within eCTD. | |
| 14.1 | <b>Demographics Data</b> | | |
| 14.1.1 | Disposition | | |
| 14.1.1.1 | Subject Enrollment and Screen Failures– Enrolled Set | IP | |
| 14.1.1.2 | Analysis Sets – Enrolled Set | IP | |
| 14.1.1.3 | Subject Disposition – Randomized Set | IP | |
| 14.1.2 | Demographics | | |
| 14.1.2.1 | Demographics – Safety Analysis Set | IP | |
| 14.1.3 | Baseline Characteristics | | |
| 14.1.3.1 | Medical History – Safety Analysis Set | IP | |
| 14.1.4.1 | Prior Medications – Safety Analysis Set | IP | |
| 14.1.4.2 | Concomitant Medications – Safety Analysis Set | IP | 14.1.4.1 |
| 14.2 | Efficacy Data | | |
| 14.2.1 | Primary Efficacy Endpoint | | |
| | Not Applicable | | |
| 14.2.2 | Secondary Efficacy Endpoints | | |
| | Not Applicable | | |
| 14.3 | Safety Data | | |
| 14.3.1 | Displays of Adverse Events | | |
| 14.3.1.1.1 | Overall Summary Adverse Events (TEAEs) by | IP | |
| | Treatment Group – Safety Analysis Set | | |
| 14.3.1.1.2 | Overall Summary Adverse Events (TEAEs) by | IP | 14.3.1.1.1 |
| | Treatment Period – Safety Analysis Set | | |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

#### **Confidentiality Statement**



Sponsor: Xeris Pharmaceuticals, Inc.

Protocol Number: DPI-201

#### STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| Table<br>Number | Table Title | Validation<br>Method | Shell<br>Number<br>(if repeat) |
|---|---|---|---|
| 14.3.1.2.1 | Any AEs by Primary System Organ Class and<br>Preferred Term by Treatment Group – Safety<br>Analysis Set | IP | |
| 14.3.1.2.2 | Any AEs by Primary System Organ Class and<br>Preferred Term by Treatment Period – Safety<br>Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.3.1 | TEAEs by Primary System Organ Class and Preferred<br>Term by Treatment Group – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.3.2 | TEAEs by Primary System Organ Class and Preferred<br>Term by Treatment Period – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.4.1 | Treatment-Related TEAEs by Primary System Organ<br>Class and Preferred Term by Treatment Group –<br>Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.4.2 | Treatment-Related TEAEs by Primary System Organ<br>Class and Preferred Term by Treatment Period –<br>Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.5.1 | Severe or Life-Threatening TEAEs by Primary System Organ Class and Preferred Term by Treatment Group – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.5.2 | Severe or Life-Threatening TEAEs by Primary System Organ Class and Preferred Term by Treatment Period – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.6.1 | Serious TEAEs by Primary System Organ Class and<br>Preferred Term by Treatment Group – Safety<br>Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.6.2 | Serious TEAEs by Primary System Organ Class and<br>Preferred Term by Treatment Period – Safety<br>Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.7.1 | Treatment-Related Serious TEAEs by Primary System Organ Class and Preferred Term by Treatment Group – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.7.2 | Treatment-Related Serious TEAEs by Primary System Organ Class and Preferred Term by Treatment Period – Safety Analysis Set | IP | 14.3.1.2.1 |

| QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 | Governing QMD: Worldwide-SOP-ST-001 |
|---|---|
|---|---|

Confidentiality Statement



Sponsor: Xeris Pharmaceuticals, Inc.

Protocol Number: DPI-201

## STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| Table<br>Number | Table Title | Validation<br>Method | Shell<br>Number<br>(if repeat) |
|---|---|---|---|
| 14.3.1.8.1 | SAEs Leading to Death by Primary System Organ<br>Class and Preferred Term by Treatment Group –<br>Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.8.2 | SAEs Leading to Death by Primary System Organ<br>Class and Preferred Term by Treatment Period –<br>Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.9.1 | TEAEs Leading to Early Withdrawal by Primary<br>System Organ Class and Preferred Term by<br>Treatment Group – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.9.2 | TEAEs Leading to Early Withdrawal by Primary<br>System Organ Class and Preferred Term by<br>Treatment Period – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.10.1 | Serious TEAEs Leading to Early Withdrawal by<br>Primary System Organ Class and Preferred Term by<br>Treatment Group – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.1.10.2 | Serious TEAEs Leading to Early Withdrawal by<br>Primary System Organ Class and Preferred Term by<br>Treatment Period – Safety Analysis Set | IP | 14.3.1.2.1 |
| 14.3.2 | Listings of Deaths, Other Serious and Significant<br>Adverse Events | | |
| 14.3.3 | Narratives of Deaths, Other Serious and Certain<br>Other Significant Adverse Events | | |
| | Not Applicable | IP | |
| 14.3.4 | Abnormal Laboratory Values | | |
| 14.3.5 | Extent of Exposure, Dosage Information, And Compliance | | |
| 14.3.5.1 | Exposure by Treatment Sequence – Safety Analysis<br>Set | IP | |
| 14.3.5.2 | Exposure by Treatment Group | IP | |
| 14.3.6 | Vital Signs and Physical Examination | | |
| 14.3.6.1.1 | Vital Signs, Descriptive Statistics and Changes from<br>Baseline to Post-Dose Assessments – Safety Analysis<br>Set | IP | |
| 14.3.6.2.1 | Physical Examination Data, Shift Table – Safety<br>Analysis Set | IP | |
| 14.3.7 | Other Safety | | |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

**Confidentiality Statement** 



Sponsor: Xeris Pharmaceuticals, Inc.

Protocol Number: DPI-201

## STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| Table<br>Number | Table Title | Validation<br>Method | Shell<br>Number<br>(if repeat) |
|---|---|---|---|
| 14.3.7.1.1 | Hematology Data, Descriptive Statistics – Safety<br>Analysis Set | IP | 14.3.6.1.1 |
| 14.3.7.1.2 | Hematology Data, Normal Range Shifts – Safety<br>Analysis Set | IP | 14.3.6.2.1 |
| 14.3.7.2.1 | Serum Chemistry Data, Descriptive Statistics – Safety<br>Analysis Set | IP | 14.3.6.1.1 |
| 14.3.7.2.2 | Serum Chemistry Data, Normal Range Shifts – Safety<br>Analysis Set | IP | 14.3.6.2.1 |
| 14.3.7.3.1 | C-Peptide and HbA1c Data, Descriptive Statistics – Safety Analysis Set | IP | 14.3.6.1.1 |
| 14.3.7.4.1 | ECG Data, Descriptive Statistics – Safety Analysis<br>Set | IP | 14.3.6.1.1 |
| 14.3.7.4.2 | ECG Data, Overall Interpretation Summary – Safety<br>Analysis Set | IP | |
| 14.3.7.5.1 | Draize Scale, Descriptive Statistics – Safety Analysis<br>Set | IP | |
| 14.3.7.6.1 | Injection Site Discomfort Assessment – Numeric<br>Rating Scale (NRS), Descriptive Statistics – Safety<br>Analysis Set | IP | 14.3.6.1.1 |
| 14.3.7.6.2 | Injection Site Discomfort Assessment – Injection Site Discomfort Description and Duration Questionnaire, Descriptive Statistics – Safety Analysis Set | IP | |
| 14.3.8.1 | Time to IV Dextrose Administration from Study Drug<br>Administration by Treatment Group – Safety<br>Analysis Set | IP | |
| 14.3.8.2 | Time to Hypoglycemic Event from Study Drug Administration by Treatment Group – Safety Analysis Set | IP | 14.3.8.1 |
| 14.3.8.3 | Time to Resolution of Hypoglycemic Event from IV Dextrose Administration by Treatment Group – Safety Analysis Set | IP | 14.3.8.1 |
| 14.3.8.4 | Proportion of Subjects Reaching Euglycemia after IV Dextrose Administration by Treatment Group – Safety Analysis Set | IP | |
| 14.3.8.5 | Average Amount of IV Dextrose by Treatment Group – Safety Analysis Set | IP | |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-ST-001

**Confidentiality Statement** 

# WORLDWIDE STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| Table<br>Number | Table Title | Validation<br>Method | Shell<br>Number<br>(if repeat) |
|---|---|---|---|
| 14.4 | PK Tables | | |
| | Separate SAP for PK analyses | | |
| 14.5 | PD Tables | | |
| 14.5.1 | Plasma Glucose Concentration Data, Descriptive | IP | 14.4.1.1 |
| | Statistics – PD Analysis Set | | |
| 14.5.2 | Plasma Glucose PD Parameter Data, Descriptive | Stat IP | 14.4.1.2 |
| | Statistics and Analysis – PD Analysis Set | | |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

**Confidentiality Statement** 



Sponsor: Xeris Pharmaceuticals, Inc.

Protocol Number: DPI-201

## STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| Figure<br>Number | Figure Title | Validation<br>Method | Shell<br>Number (if<br>repeat) |
|---|---|---|---|
| 14.3.1.1 | Time to IV Dextrose Administration from Study Drug<br>Administration by Treatment Group – Safety Analysis<br>Set | IP | |
| 14.3.1.2 | Time to Hypoglycemic Event from Study Drug<br>Administration by Treatment Group—Safety Analysis<br>Set | IP | 14.3.1.1 |
| 14.3.1.3 | Time to Resolution of Hypoglycemic Event from IV Dextrose Administration by Treatment Group—Safety Analysis Set | IP | 14.3.1.1 |
| 14.5.1.1 | Plasma Glucose Concentration Data, Mean Profiles on<br>Linear Scale – PD Analysis Set | IP | |
| 14.5.1.2 | Plasma Glucose Concentration Data, Individual Profiles<br>on Linear Scale – PD Analysis Set | IP | |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001



Sponsor: Xeris Pharmaceuticals, Inc.

Protocol Number: DPI-201

## STATISTICAL ANALYSIS PLAN. PHASE 2-3-4

| Listing<br>Number | Listing Title | Validation<br>Method | Shell<br>Number<br>(if repeat) |
|---|---|---|---|
| 16.2 | Subject Data Listings | | |
| 16.2.1 | Discontinued Subjects | | |
| 16.2.1.1 | Screen Failures – Enrolled Set | IP | |
| 16.2.1.2 | Inclusion/Exclusion Criteria – Enrolled Set | IP | |
| 16.2.1.3 | Study Completion – Safety Analysis Set | IP | |
| 16.2.2 | Protocol Deviations | | |
| 16.2.2.1 | Protocol Deviations – Enrolled Set | IP | |
| 16.2.3 | Subjects Excluded from the Efficacy Analyses | | |
| 16.2.3.1 | Analysis Sets – Enrolled Set | IP | |
| 16.2.4 | Demographic Data | | |
| 16.2.4.1 | Demographic Data – Safety Analysis Set | IP | |
| 16.2.4.2 | Medical History – Safety Analysis Set | IP | |
| 16.2.4.2 | Prior/Concomitant Medications – Safety Analysis Set | IP | |
| 16.2.5 | Compliance and / or Drug Concentration Data | | |
| 16.2.5.1.1 | Exposure – Safety Analysis Set | IP | |
| 16.2.6 | Individual Efficacy Response Data | | |
| | Not Applicable | | |
| 16.2.7 | Adverse Event Listings | | |
| 16.2.7.1 | Adverse Events – Safety Analysis Set | IP | |
| 16.2.8 | Individual Laboratory Measurements and Other Safety | | |
| 16.2.8.1.1 | Vital Sign Data – Safety Analysis Set | IP | |
| 16.2.8.2.1 | Physical Examination Data – Safety Analysis Set | IP | |
| 16.2.8.3.1 | Hematology Data – Safety Analysis Set | IP | |
| 16.2.8.3.2 | Serum Chemistry Data – Safety Analysis Set | IP | |
| 16.2.8.3.3 | C-Peptide and HbA1c Data – Safety Analysis Set | IP | |
| 16.2.8.3.4 | Urine Drug Screen Data – Safety Analysis Set | IP | |
| 16.2.8.3.5 | Urine Pregnancy Test Data – Safety Analysis Set | IP | |
| 16.2.8.4.1 | ECG Data – Safety Analysis Set | IP | |
| 16.2.8.5.1 | Draize Scale Data – Safety Analysis Set | IP | |
| 16.2.8.6.1 | Injection Site Discomfort Assessment Data – Safety<br>Analysis Set | IP | |
| 16.2.8.7.1 | Plasma Glucose Concentration Data, Descriptive<br>Statistics – Safety Analysis Set | IP | |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019 Governing QMD: Worldwide-SOP-ST-001

**Confidentiality Statement**
#### WORLDWIDE STATISTICAL ANALYSIS PLAN. PHASE 2-3-4 Worldwide Clinical Trials Controlled Quality Management Document Sponsor: Xeris Pharmaceuticals, Inc. DPI-201

| Listing<br>Number | Listing Title | Validation<br>Method | Shell<br>Number<br>(if repeat) |
|---|---|---|---|
| 16.2.8.7.2 | Plasma Glucose PD Parameter Data – Safety Analysis | IP | |
| | Set | | |
| 16.2.8.7.3 | Glucose Challenge – Safety Analysis Set | IP | |
| 16.2.8.8.1 | Hypoglycemic Events – Safety Analysis Set | IP | |

QMD Ref: Worldwide-TMP-ST-005-7.0 Effective: 12Aug2019

Governing QMD: Worldwide-SOP-ST-001

This document is the property of Worldwide Clinical Trials Inc. and may not be duplicated, copied, altered or removed from company without prior approval from Worldwide Quality Assurance or in compliance with Worldwide Standard Operating Procedures.

Page X of Y

Table 14.1.1.1 Subject Enrollment and Screen Failures Enrolled Set

| | Overall |
|-------------------------------|------------------|
| | (N=XXX)<br>n (%) |
| Number of Subjects Enrolled | xx (xx.x) |
| Site | |
| Site 1 | xx (xx.x) |
| Site 2 | XX (XX.X) |
| Site 3 | xx (xx.x) |
| | xx (xx.x) |
| Number of Screen Failures | xx (xx.x) |
| Reason for Screen Failure (a) | |
| Reason 1 | xx (xx.x) |
| Reason 2 | xx (xx.x) |
| Reason 3 | xx (xx.x) |
| | xx (xx.x) |

PROGRAMMING NOTE: Reasons: 'Withdrawal of Consent', 'Did Not Meet Inclusion/Exclusion Criteria', 'Adverse Event', 'Lost to Follow-Up', 'Pregnancy', 'Other'.

Worldwide Clinical Trials DDMMMYYYY:HH:MM

| | | | B-A-C | (N=XXX) |
|----------------|---------------|--------------|-------|---------|
| | | | A-C-B | (N=XXX) |
| Table 14.1.1.2 | Analysis Sets | Enrolled Set | C-A-B | (N=XXX) |
| | | | B-C-A | (N=xxx) |
| | | | A-B-C | (N=XXX) |

| Analysis Set | A-B-C<br>(N=xxx)<br>n (%) | B-C-A<br>(N=xxx)<br>n (%) | C-A-B<br>(N=xxx)<br>n (%) | A-C-B<br>(N=xxx)<br>n (%) | B-A-C<br>(N=xxx)<br>n (%) | C-B-A<br>(N=xxx)<br>n (%) | Overall (N=xxx) n (%) |
|---|---|---|---|---|---|---|---|
| Analysis Set 1 | (x.xx) xx | xx (xx.x) | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx | xx (xx.x) |
| Analysis Set 2 | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Analysis Set 3 | xx (xx.x) | xx (xx.x) | XX (XX.X) | (xxxx) xx | (xxxx) xx | (xx.x) | (xxxx) xx |
| | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx | (xx.x) | (x.xx) xx | (x.xx) |

PROGRAMMING NOTE: Use analysis sets: 'Enrolled Set', 'Randomized Set', 'Safety Analysis Set', 'PD Analysis Set'.

PROGRAMMING NOTE: Do not display treatment sequence frequencies for 'Enrolled Set' where only overall should be displayed.

Randomized Set: All subjects who were randomized to the treatment sequence.

Safety Analysis Set: All randomized subjects who received any study drug.

PD Analysis Set: Subset of the Safety Analysis Set, which includes subjects who had blood glucose measured at pre-dose and 180 minutes post-dose, and at least one time point between pre-dose and 180 minutes post-dose.

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.1.1.3 Subject Disposition Randomized Set


| Disposition | A-B-C<br>(N=xxx)<br>n (%) | B-C-A<br>(N=xxx)<br>n (%) | C-A-B<br>(N=xxx)<br>n (%) | A-C-B<br>(N=xxx)<br>n (%) | B-A-C<br>(N=xxx)<br>n (%) | C-B-A<br>(N=xxx)<br>n (%) | Overall (N=xxx) n (%) |
|---|---|---|---|---|---|---|---|
| Completed Study (a) | (xx.x) | (x.x.) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x · xx) xx | xx (xx.x) |
| Early Withdrawal (a) | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx | (xx) xx | (x.xx) xx | (x.x.x) |
| Primary Reason for Early Withdrawal (b) | | | ( > | (> >> | (\$ \$\$) | ( > | (>>>) |
| Reason 2 | | (x.xx) xx | (x.xx) xx | (x:xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx |
| Reason 3 | (xx) | (x.xx) xx | (xx.x) xx | (x.xx) xx | (xx.xx) xx | (x.xx) xx | (xx.x) |
| : | (x.xx) xx | xx (xx.x) | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx | xx (xx.x) |
| Time to Early Withdrawal (days) | | | | | | | |
| n | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| Mean (SD) | xx.xx) x.xx | xx.xx (xx.xx) | xx.x (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | ×. ×. | xx.xx | ×.×. | x.x. | ××.× | x.xx | x.xx |
| Min, Max | xx 'xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

PROGRAMMING NOTE: Reasons: 'Withdrawal of Consent', 'Did Not Meet Inclusion/Exclusion Criteria', 'Adverse Event', 'Lost to Follow-Up', 'Pregnancy', 'Other'.

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.1.2.1 Demographics


Safety Analysis Set

| Parameter | A-B-C<br>(N=xxx) | B-C-A<br>(N=xxx) | C-A-B<br>(N=xxx) | A-C-B<br>(N=xxx) | B-A-C<br>(N=XXX) | C-B-A<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|---|---|---|
| Categorical Variable 1, n (%) | | | | | | | |
| Category 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Category 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Category 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| : | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Continuous Variable 1 (unit) | | | | | | | |
| n | ×× | ×× | XX | ×× | ×× | ×× | XX |
| Mean (SD) | xx.xx (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.xx) xxxx | xx.x (xx.xx) | xx.xx) xxxx |
| Median | ×.×. | x.xx | x.x. | xx.x | xx.x | ×. ×× | xx.x |
| Min, Max | xx, xx | xx, xx | xx 'xx | xx, xx | xx, xx | xx, xx | xx, xx |

PROGRAMMING NOTE: Age (years), Gender ('Male', 'Female'), Childbearing Potential ('Yes', 'No'), Ethnicity ('Hispanic or Latino', 'Not Hispanic or Latino'), Race ('White', 'Black or African American', 'Asian', 'American Indian or Alaska Native', 'Native Hawaiian or Other Pacific Islander', 'Multiple'), Weight (kg), Height (cm) and Body Mass Index (kg/m2).

Program: XXX.SAS


Table 14.1.3.1 Medical History Safety Analysis Set

| System Organ Class<br>Preferred Term | A-B-C (N=xxx) n (%) / Events | B-C-A<br>(N=xxx)<br>n (%) / Events | C-A-B<br>(N=xxx)<br>n (%) / Events | A-C-B<br>(N=xxx)<br>n (%) / Events | B-A-C (N=xxx) n (%) / Events | C-B-A<br>(N=xxx)<br>n (%) / Events | Overall (N=xxx) n (%) / Events |
|---|---|---|---|---|---|---|---|
| Any | xx / (x.xx) xx | xx / (x.xx) xx | xx / (xx.x) / xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| System Organ Class 1<br>Preferred Term 1 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx xx / (x.xx) xx | xx / (x.xx) xx x / (x.xx) xx x / (x.xx) x x / (x.xx) x / (x | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 2 | xx / (xx.xx) xx | xx / (xx.xx) xx | xx / (xx.xx) xx | xx / (x.xx) xx | xx / (xx.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 3 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| : | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| System Organ Class 2 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (xxxx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 1 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 2 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 3 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| ÷ | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | | xx / (x.xx) xx xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |

## PROGRAMMING NOTE:


Table 14.1.4.1 Prior Medications Safety Analysis Set

| | A-B-C | B-C-A | C-A-B | A-C-B | B-A-C | C-B-A | Overall |
|---|---|---|---|---|---|---|---|
| ATC Level 4 | (N=xxx) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=xxx) | (N=XXX) |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Any | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) xx | xx (xx.x) |
| ATC Class 1 | (x.xx) | (x.xx) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | (x.xx) xx | (xxxx) xx | xx (xx.x) | (xxxx) xx | xx (xx.x) | xx (xx.x) | (xxxx) xx |
| Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| : | (x.xx) | (x.xx) xx | xx (xx.x) | (x.xx) xx | (x.x.x) xx | (x.xx) xx | (x.xx) xx |
| ATC Class 2 | (x.xx) | (x.xx) xx | xx (xx.x) | (x.xx) xx | (xx.x) | (x.xx) xx | (xxx) xx |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xxxx) xx |
| Preferred Term 3 | (x.xx) xx | (xxxx) xx | xx (xx.x) | (xxxx) xx | xx (xx.x) | xx (xx.x) | (xxxx) xx |
| :: | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) | xx (xx.x) | (xx.x) | xx (xx.x) |

# PROGRAMMING NOTE:

Worldwide Clinical Trials DDMMMYYYY:HH:MM

PROGRAMMING NOTE: Same shell as Table 14.1.4.1.

Xeris Pharmaceuticals, Inc. DPI-201

Overall Summary of Adverse Events by Treatment Group Safety Analysis Set Table 14.3.1.1.1

| AE Category | XP-39249<br>(N=xxx)<br>n (%) / Events | Regular Insulin (N=xxx) n (%) / Events | Regular Insulin + Pramlintide (N=xxx) n (%) / Events | Overall (N=xxx) n (%) / Events |
|---|---|---|---|---|
| Category 1 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (xx.x) xx |
| Category 2 | xx / (xx.x) xx | xx / (x.xx) xx | xx / (xx.x) xx | xx / (x.xx) xx |
| Category 3 | xx / (xx.x) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (xxxx) xx |
| | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |

PROGRAMMING NOTE: Include AE Categories: 'Any AEs', 'Teatment-Related TEAEs', 'Severe or Life-Threatening TEAEs', 'Serious TEAEs', 'Treatment-Related Serious TEAEs', 'SAEs Leading to Death', 'TEAEs Leading to Early Withdrawal', 'Serious TEAEs Leading to Early Withdrawal', 'Serious TEAEs', 'SAEs Leading to Death', 'TEAEs Leading to Early Withdrawal', 'Serious TEAEs', 'SAEs Leading to Death', 'TEAEs Leading to Early Withdrawal', 'Serious TEAEs Leading to Early Withdrawal', 'Serious TEAEs', 'Severe or Life-Threatening TEAEs', 'Serious TEAEs', 'Treatment-Related TEAEs', 'Serious TE

TEAE = Treatment-Emergent Adverse Event.

Program: XXX.SAS

Table 14.3.1.1.2 Overall Summary of Adverse Events by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.1.1 using Treatment Period instead of Treatment Group.

Page X of Y

Table 14.3.1.2.1 Any AEs by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

| System Organ Class<br>Preferred Term | XP-3924<br>(N=xxx)<br>n (%) / Events | Regular Insulin<br>(N=xxx)<br>n (%) / Events | Regular Insulin + Pramlintide (N=xxx) n (%) / Events | Overall (N=xxx) n (%) / Events |
|---|---|---|---|---|
| Any | xx / (xx.x) xx | xx / (xx.x) xx | xx / (x.x.) xx | xx / (x.xx) xx |
| System Organ Class 1 | | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 1<br>Preferred Term 2 | xx (xx.x) / xx<br>xx (xx.x) / xx | xx / (x.xx) xx<br>xx / (x.xx) xx | xx (xx.x) / xx<br>xx (xx.x) / xx | xx (xx.x) / xx<br>xx (xx.x) / xx |
| Preferred Term 3 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| ÷ | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| System Organ Class 2 | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 1 | xx / (xx.x) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| Preferred Term 2 | xx / (xx.x) xx | xx / (xxxx) xx | xx / (x.xx) xx | xx / (xxxx) xx |
| Preferred Term 3 | xx / (xx.x) xx | xx / (x.xx) xx | xx / (x.xx) xx | xx / (x.xx) xx |
| :: | xx / (xxxx) xx | xx / (x.xx) xx | xx / (x.x.) xx | xx / (x.xx) xx |

### PROGRAMMING NOTE:

Table 14.3.1.2.2 Any AEs by Primary System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.2.1 using Treatment Period instead of Treatment Group.

Page X of Y

TEAEs by System Organ Class and Preferred Term by Treatment Group Safety Analysis Set Table 14.3.1.3.1

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

Table 14.3.1.3.2 TEAEs by System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.3.1 using Treatment Period instead of Treatment Group.

Table 14.3.1.4.1 Treatment-Related TEAEs by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

Table 14.3.1.4.2

Treatment-Related TEAEs by Primary System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.4.1 using Treatment Period instead of Treatment Group.

Program: XXX.SAS

Table 14.3.1.5.1 Severe or Life-Threatening TEAEs by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

Table 14.3.1.5.2 Severe or Life-Threatening TEAEs by Primary System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.5.1 using Treatment Period instead of Treatment Group.

Table 14.3.1.6.1 Serious TEAEs by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

n = Number of subjects with event, Events = Total number of events. Adverse events are coded using MedDRA version 22.0. TEAE = Treatment-Emergent Adverse Event.

Program: XXX.SAS

PROGRAMMING NOTE: Repeat Table 14.3.1.6.1 using Treatment Period instead of Treatment Group.

Table 14.3.1.7.1 Treatment-Related Serious TEAEs by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

Treatment-Related Serious TEAEs by Primary System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.7.1 using Treatment Period instead of Treatment Group.

Table 14.3.1.8.1 SAEs Leading to Death by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

Table 14.3.1.8.2 SAEs Leading to Death by Primary System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.8.1 using Treatment Period instead of Treatment Group.

TEAES Leading to Early Withdrawal by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

Table 14.3.1.9.2 TEAEs Leading to Early Withdrawal by Primary System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.9.1 using Treatment Period instead of Treatment Group.

Table 14.3.1.10.1 Serious TEAEs Leading to Early Withdrawal by Primary System Organ Class and Preferred Term by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.1.2.1.

Table 14.3.1.10.2 Serious TEAEs Leading to Early Withdrawal by Primary System Organ Class and Preferred Term by Treatment Period Safety Analysis Set

PROGRAMMING NOTE: Repeat Table 14.3.1.10.1 using Treatment Period instead of Treatment Group.

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.3.5.1
Exposure by Treatment Sequence Safety Analysis Set


| Exposure | A-B-C<br>(N=xxx)<br>n (%) | B-C-A<br>(N=xxx)<br>n (%) | C-A-B<br>(N=xxx)<br>n (%) | A-C-B<br>(N=xxx)<br>n (%) | B-A-C<br>(N=xxx)<br>n (%) | C-B-A<br>(N=xxx)<br>n (%) | Overall (N=xxx) n (%) |
|---|---|---|---|---|---|---|---|
| Subjects with 3 treatments Subjects with 2 treatments Subjects with 1 treatments Subjects with 0 treatments | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with Period 1 treatment | xx (xx.x) | xx (xx.x) | ×× | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with Period 2 treatment | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with Period 3 treatment | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

# PROGRAMMING NOTE:

Table 14.3.5.2 Exposure by Treatment Group Safety Analysis Set

| | S S S S S S S S S S S S S S S S S S S | Regular Insulin + Pramlintide (N=xxx) n (%) | Overall (N=xxx) n (%) |
|---|---|---|---|
| NullDet Of SUDJECTS treated | (v.v.) vv (v. | (****) ** | (x.xx) xx |

# PROGRAMMING NOTE:

Program: XXX.SAS

Table 14.3.6.1.1 Vital Signs, Descriptive Statistics and Changes from Baseline to Post-Dose Assessments Safety Analysis Set

Parameter: XXX (Unit)

| Treatment | Visit | Timepoint | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|
| XP-3924 (N=xxx) | Visit 1 | Observed value | ×× | x.xx | xx · xx | x.xx | ×× | ×× |
| | Visit 2<br>Visit 2 | Observed value<br>Change from BL | × × | × | xx.xx<br>xx.xx | × | × ×<br>× × | × ×<br>× × |
| | Visit 3<br>Visit 3 | Observed value<br>Change from BL | × ×<br>× × | × | xx.xx<br>xx.xx | × | × × | × ×<br>× × |
| | : : | Observed value<br>Change from BL | × ×<br>× × | × | ××.××<br>××.×× | × ×<br>× ×<br>× × | × ×<br>× × | × ×<br>× × |
| Regular Insulin<br>(N=xxx) | Visit 1 | Observed value | ×× | × × × × | ×× · ×× | x . x x | ×× | ×× |
| | Visit 2<br>Visit 2 | Observed value<br>Change from BL | × ×<br>× × | × × × × × | ××.××<br>××.×× | × × × × × | × × | × ×<br>× × |
| | Visit 3<br>Visit 3 | Observed value<br>Change from BL | × × | ×: ×:<br>× ×: | ×× · × | × | × ×<br>× × | × ×<br>× × |
| | : : | Observed value<br>Change from BL | × ×<br>× × | × · × | ××.××<br>××.×× | x x x x x x x x x x x x x x x x x x x | × ×<br>× × | × ×<br>× × |
| Regular Insulin +<br>Pramlintide (N=xxx) | Visit 1 | Observed value | ×× | ×·×× | ××·×× | ×·×× | ×× | × |
| | Visit 2<br>Visit 2 | Observed value<br>Change from BL | × × | × × × × × | xx · xx<br>xx · xx | × | × ×<br>× × | × ×<br>× × |
| | Visit 3<br>Visit 3 | Observed value<br>Change from BL | × ×<br>× × | × ×<br>× ×<br>× × | xx · xx<br>x · xx | × ×<br>× × | × ×<br>× × | × ×<br>× × |
| | : | Observed value | XX | ×× | XX.XX | xx.x | ×× | XX |

Page X of Y

Table 14.3.6.1.1

Vital Signs, Descriptive Statistics and Changes from Baseline to Post-Dose Assessments Safety Analysis Set

Parameter: XXX (Unit)

| Treatment | Visit | Timepoint | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|
| | : | Change from BL | XX | ×·×× | ××.×× | × · ×× | ×× | ×× |
| Overall (N=xxx) | Visit 1 | Observed value | ×× | X. XX | xx.xx | x · xx | ×× | ×× |
| | Visit 2 | Observed value | ×× | ×. ×× | ××.×× | x. xx | ×× | ×× |
| | Visit 2 | Change from BL | ×× | ×. ×× | xx.xx | xx | ×× | ×× |
| | Visit 3 | Observed value | ×× | ×.×× | ××.×× | x. xx | ×× | ×× |
| | Visit 3 | Change from BL | ×× | ×. ×× | xx.xx | x. xx | ×× | ×× |
| | : | Observed value | ×× | × · × × | ××. ×× | x.xx | ×× | ×× |
| | : | Change from BL | ×× | ×× | XX.XX | xx.x | ×× | ×× |

PROGRAMMING NOTE: For each treatment group include following visits: 'Pre-Dose', '30 min Post-Dose', '180 min Post-Dose', '360 min Post-Dose'.

PROGRAMMING NOTE: For overall treatment group include following visits: 'Screening', 'Follow-Up'.

Xeris Pharmaceuticals, Inc. DPI-201


Table 14.3.6.2.1 Physical Examination Data, Shift Table Safety Analysis Set

Parameter: XXX (Unit)

| | | | | Follow-Up | | |
|---|---|---|---|---|---|---|
| Treatment | Screening | Normal | Abnormal (NCS) | Abnormal (CS) | Not Done | Overall |
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Overall (N=xxx) | Normal | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Overall (N=xxx) | Abnormal (NCS) | XX (XX.X) | xx (xx.x) | xx (xx.x) | (xx.x) xx | (x.xx) xx |
| Overall (N=xxx) | Abnormal (CS) | XX (XX.X) | (xx.x) xx | xx (xx.x) | (xxxx) xx | xx (xx.x) |
| Overall (N=xxx) | Not Done | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) xx | xx (xx.x) |
| Overall (N=xxx) | Overall | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

PROGRAMMING NOTE: Percentages are based on number of subjects who had both Screening and Follow-up records.

Worldwide Clinical Trials DDMMMYYYY:HH:MM

Table 14.3.7.1.1
Hematology Data, Descriptive Statistics
Safety Analysis Set

Parameter: XXX (Unit)

PROGRAMMING NOTE: Same shell as Table 14.3.6.1.1 including only overall treatment and visits 'Screening', 'Follow-Up'.

PROGRAMMING NOTE: Include parameters as listed in the Protocol.

PROGRAMMING NOTE: Same shell as Table 14.3.6.2.1 using categories 'Low', 'Normal', 'High', 'Overall'.

PROGRAMMING NOTE: Include parameters as listed in the Protocol.

PROGRAMMING NOTE: Percentages are based on number of subjects who had both Screening and Follow-up records.

Page X of Y

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.3.7.2.1 Serum Chemistry Data, Descriptive Statistics Safety Analysis Set

Parameter: XXX (Unit)

PROGRAMMING NOTE: Same shell as Table 14.3.6.1.1 including only overall treatment and visits 'Screening', 'Follow-Up'.

PROGRAMMING NOTE: Include parameters as listed in the Protocol.

Worldwide Clinical Trials DDMMMYYYY:HH:MM Program: XXX.SAS
PROGRAMMING NOTE: Same shell as Table 14.3.6.2.1 using categories 'Low', 'Normal', 'High', 'Overall'.

PROGRAMMING NOTE: Include parameters as listed in the Protocol.

PROGRAMMING NOTE: Percentages are based on number of subjects who had both Screening and Follow-up records.

Table 14.3.7.3.1 C-Peptide and HbAlc Data, Descriptive Statistics Safety Analysis Set

Parameter: XXX (Unit)

PROGRAMMING NOTE: Same shell as Table 14.3.6.1.1 including only overall treatment and visit 'Screening'.

Worldwide Clinical Trials DDMMMYYYY:HH:MM Program: XXX.SAS

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.3.7.4.1 ECG Data, Descriptive Statistics Safety Analysis Set

Parameter: XXX (Unit)

PROGRAMMING NOTE: Same shell as Table 14.3.6.1.1 including only overall treatment and visit 'Screening'.

Worldwide Clinical Trials DDMMMYYYY:HH:MM Program: XXX.SAS

Table 14.3.7.4.2 ECG Data, Overall Interpretation Summary Safety Analysis Set

| Overall (N=xxx) Result n (%) | Normal Abnormal NCS Abnormal CS Abnormal C |
|---|---|
| Parameter | XXX (Unit) XXX (Unit) XXX (Unit) |

PROGRAMMING NOTE: Including only visit 'Screening'.

PROGRAMMING NOTE: Percentages are based on number of subjects who had record at the visit.

Draize Scale, Descriptive Statistics Safety Analysis Set Table 14.3.7.5.1

Page X of Y

Parameter: XXX (Unit)

| Timepoint | Result | XP-3924<br>(N=xxx)<br>n (%) | Regular Insulin (N=xxx) n (%) | Regular Insulin + Pramlintide (N=xxx) n (%) | Overall (N=xxx) n (%) |
|---|---|---|---|---|---|
| XXX<br>XXX | Result 1<br>Result 2<br>Result 2 | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

PROGRAMMING NOTE: Erythema Formation: '0 - No erythema', '1 - Very slight erythema', '2 - Well defined erythema', '3 - Moderate erythema', '4 - Severe erythema'.

PROGRAMMING NOTE: Edema Formation: '0 - No edema', '1 - Very slight edema', '2 - Well defined edema', '3 - Moderate edema'.

PROGRAMMING NOTE: Including timepoints '30 min Post-Dose', '90 min Post-Dose', '360 min Post-Dose'.

PROGRAMMING NOTE: Percentages are based on number of subjects who had record at the timepoint.

Table 14.3.7.6.1 Injection Site Discomfort Assessment - Numeric Rating Scale (NRS), Descriptive Statistics Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.6.1.1 not having change from BL. Use 'Timepoint' Instead of 'Visit'.

PROGRAMMING NOTE: Including timepoints '10 min Post-Dose', '30 min Post-Dose'.

PROGRAMMING NOTE: Percentages are based on number of subjects who had record at the timepoint.

Injection Site Discomfort Assessment - Injection Site Discomfort Description and Duration Questionnaire, Descriptive Statistics Safety Analysis Set Table 14.3.7.6.2

| Result | XP-3924<br>(N=xxx) | Regular Insulin<br>(N=xxx) | Regular Insulin + Pramlintide (N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|
| How would you describe any discomfort you felt from the study drug? n (%) | from the study drug? n (%) | | | |
| None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Itching | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tingling, twitching, or numbness | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Irritation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| About how long did the discomfort last after the injection? n | e injection? n (%) | | | |
| Less than 1 minute | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1-2 minutes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3-5 minutes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6-9 minutes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At least 10 minutes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| In total, how long did the discomfort last after the injection? (minutes) | r the injection? (minutes) | | | |
| ч | ×× | ×× | ×× | ×× |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | x.x.x | xx.xx | x.xx | ×.×. |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |

PROGRAMMING NOTE: Percentages are based on number of subjects who had study treatment. Add missing categories if needed.

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.3.8.1 Time (minutes) to IV Dextrose Administration from Study Drug Administration by Treatment Group Safety Analysis Set

| | XP-3924<br>(N=xxx) | Regular Insulin | Regular Insulin + Pramlintide (N=xxx) |
|---|---|---|---|
| Number (%) of Subjects with Event<br>Number (%) of Subjects Censored | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Kaplan-Meier estimates (95% CI) | | | |
| 25th percentile | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Median | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| 75th percentile | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Log-Rank | | | |
| Chi-Square (DF) | xx.xx (x) | xx.xx (x) | xx.xx (x) |
| p-value | x.xx | x.xxx | X.XXX |
| Mean Time (min) (SE) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

Table 14.3.8.2 Time (minutes) to Hypoglycemic Event from Study Drug Administration by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.8.1.

If hypo event occurs after glucose challenge then it will not be included as event and will be censored at the time of glucose challenge. Only events occurring after treatment and prior to glucose challenge are included as events.

Program: XXX.SAS

Table 14.3.8.3 Time (minutes) to Resolution of Hypoglycemic Event from IV Dextrose Administration by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Table 14.3.8.1.

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.3.8.4 Proportion of Subjects Reaching Euglycemia after IV Dextrose Administration by Treatment Group Safety Analysis Set

| Timepoint | XP-3924<br>(N=xxx)<br>n / f (%) | Regular Insulin<br>(N=xxx)<br>n / f (%) | Regular Insulin + Pramlintide (N=xxx) n / f (%) |
|---|---|---|---|
| XXX | xx / xx (xx.x) | xx / xx (xx.x) | xx / xx (xx.x) |
| XXX | xx / xx (xx.x) | xx / xx (xx.x) | xx / xx (xx.x) |
| XXX | xx / xx (xx.x) | xx / xx (xx.x) | xx / xx (xx.x) |

PROGRAMMING NOTE: Including timepoints '10 min', '20 min', '30 min'.

# PROGRAMMING NOTE:


Table 14.3.8.5

Average Amount of IV Dextrose (g) by Treatment Group
Safety Analysis Set

| XP-3924 (N=xxx) xx xx.xx | Max | 01 03 | 95% CI | %CA |
|---|---|---|---|---|
| xxxx xxxxx xxxx xxxx + xxxxx xxxx xxxx | × | *** | (×: ×× ,×: ××) | ××× |
| ***** ***** ***** ***** ***** | | | (x.x, x.xx) | ×.× |
| XXXXX XXXXXX XXXXX | | | | |
| Framiintide (N=XXX) | × | x.xx x.xx | (XXX, XXX) | ×.<br>×× |

| Treatment Comparison | Mean | SE | 95% CI | p-value |
|---|---|---|---|---|
| XP-3924 vs. Regular Insulin | XX.XX | xx.xxx | (xx.xx, xx.xx) | XXXX.X |
| XP-3924 vs. Regular Insulin +<br>Pramlintide | XX.XX | XX.XX | (xx.xx, xx.xx) | x.xx. |
| Regular Insulin vs. Regular Insulin<br>+ Pramlintide | xx · xx | xxxx | (xx.xx, xx.xx) | × × × × |

Page X of Y

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.5.1 Plasma Glucose Concentration Data, Descriptive Statistics PD Analysis Set

Parameter: XXX (Unit)

| Treatment | Timepoint | n | Mean | SD | Median | Min | Max | 21 | 03 | 95% CI | %CV |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XP-3924 (N=xxx) | Timepoint 1 | × | ×.<br>×× | ××.<br>×× | ×.<br>×. | × | × | ×××× | ×.<br>×× | (XX.X, XX.X) | ×<br>×<br>× |
| XP-3924 (N=xxx) | Timepoint 2 | × | ×. × | ××.×× | ××.× | × | × | ×. × | xx.x | (xx.x, xx.x) | ××.× |
| XP-3924 (N=xxx) | Timepoint 3 | ×× | ×. × | ××.×× | ×. ×. | × | × | ×.× | ×. × | (xx.x, xx.x) | ××. |
| XP-3924 (N=xxx) | : | × | ×.× | ××. ×× | × × × | × | × | ×. ×. | ×.<br>×. | (xx.x, xx.x) | ×. × |
| Regular Insulin (N=xxx) | Timepoint 1 | ×× | × × × | ×× · ×× | × × × | × | × | ×.<br>×. | × × × | (x.x, xx.x) | ×. × |
| Regular Insulin (N=xxx) | Timepoint 2 | × | × × × | ××. ×× | x · xx | × | × | ×. ×× | ×.<br>×. | (xxx, xx,x) | × |
| Regular Insulin (N=xxx) | Timepoint 3 | ×× | × × × | ×× · · × | ×××× | ×× | × | × × × | ×. × | (x.x, xx.x) | ×. ×× |
| Regular Insulin<br>(N=xxx) | <u>:</u> | ×× | × | xx.xx | x.xx | × | × | × × × | × | (xxx, xxxx) | × × × |
| Regular Insulin + Pramlintide (N=xxx) | Timepoint 1 | × | × × × | ××.×× | ××× | × | × | × × × | ×<br>×<br>× | (x.x, xx.x) | ×.<br>× |
| Regular Insulin + Pramlintide (N=xxx) | Timepoint 2 | ×× | × × × | ×× · ×× | × | ×× | × | ×. ×× | ×. × | (x.xx, xx.x) | ××. |
| Regular Insulin + Pramlintide (N=xxx) | Timepoint 3 | ×× | × × × | ×× · × | ××× | ×× | × | × × × | ×. × | (x.x, xx.x) | ×. ×. |
| Regular Insulin +<br>Pramlintide (N=xxx) | ÷ | × | ×. | ×<br>×<br>× | ×· | × | × | ×<br>× | × | (xx.x, xx.x) | ××× |
| Overall (N=xxx) | Timepoint 1 | ×× | x.xx | xx.xx | ×.× | ×× | × | ××.× | × × × | (xxx, xxx) | ×. × |
| Overall (N=xxx) | Timepoint 2 | XX | ××.× | XX.XX | ×. × | ×× | XX | ×. × | ××.× | (xx,x,x,x) | ××.× |
| Overall (N=xxx) | Timepoint 3 | ×× | ××× | xx.xx | ×. ×. | × | × | ×.× | ×. × | (xx.x, xx.x) | × × × |
| Overall (N=xxx) | : | × | × | xx.xx | × . × × | × | × | x. xx | × × × | (xxx, xx.x) | ××. |

PROGRAMMING NOTE: Timepoints: 'Pre-Dose', '10 min', '20 min', '30 min', '40 min', '50 min', '60 min', '90 min', '120 min', '180 min'.

Xeris Pharmaceuticals, Inc. DPI-201

Table 14.5.2 Plasma Glucose PD Parameter Data, Descriptive Statistics and Analysis PD Analysis Set

Parameter: XXX (Unit)

| Treatment | u | n Mean | SD | SD Median | Min | Max | 21 | 03 | 95% CI | %CA |
|---|---|---|---|---|---|---|---|---|---|---|
| XP-3924 (N=xxx) | × | ××.×× | xx.xx | ××. | × | × | ××. | ××. | (xx.x, xx.x) | ×.<br>×× |
| Regular Insulin<br>(N=xxx) | × | XX.XX | XX.XX | ×.× | XX | XX | ×. × | × | (xxx, xx.x) | x. x. |
| Regular Insulin +<br>Pramlintide (N=xxx) | × | XX.X | xx · xx | ×.× | XX | ×× | x . x x | xx. | (xx.x, xx.x) | xx.x |

| Effect | Degrees of Freedom | Error Degrees of<br>Freedom | F-Statistic | p-value |
|---|---|---|---|---|
| Sequence | ×.×× | ×.×× | XX.XX | x.xx |
| Period | ×.×× | XX.X | xx.xx | X.XXX |
| Treatment | ×·×× | ××.× | xx.xx | x.xx |

Table 14.5.2 Plasma Glucose PD Parameter Data, Descriptive Statistics and Analysis PD Analysis Set

Parameter: XXX (Unit)

| Treatment | LS Mean | SE | 95% CI | p-value |
|---|---|---|---|---|
| XP-3924<br>Regular Insulin<br>Regular Insulin + Pramlintide | XX.XX<br>XX.XX<br>XX.XX | XX.XXX<br>XX.XXX | (xx.xx, xx.xx)<br>(xx.xx, xx.xx)<br>(xx.xx, xx.xx) | × |
| Treatment Comparison | LS Mean | SE | 95% CI | p-value |
| XP-3924 vs. Regular Insulin | XX.XX | XX.XX | (XX.XX, XX.XX) | x.xx |
| XP-3924 vs. Regular Insulin +<br>Pramlintide | xx.xx | xx.xx | (xx.xx, xx.xx) | x.xx.x |
| Regular Insulin vs. Regular Insulin +<br>Pramlintide | xx.xx | xxxxx | (xx.xx, xx.xx) | x.xx |

PROGRAMMING NOTE: Include parameters as specified in the Statistical Analysis Plan.

PROGRAMMING NOTE: Parameter 'Plasma glucose Tmax' is analysed using Wilcoxon Signed Rank Test so output will not have ANOVA type 3 tests or LS means. Only p-values for pairwise comparisons are displayed.

PROGRAMMING NOTE: Parameter 'Tmax' is analysed using Wilcoxon Signed Rank Test so output will not have ANOVA type 3 tests or LS means. Only p-values for pairwise comparisons are displayed.

Listing 16.2.1.1 Screen Failures Enrolled Set


| Subject Number Date | Date | Reason / | Other Reason |
|---|---|---|---|
| 12345 | DDMMMYYYY | Reason Text | Other Reason Specification Text |
| 23456 | DDMMXXXX | Reason Text | Other Reason Specification Text |
| 34567 | DDMMXXXX | Reason Text | Other Reason Specification Text |
| : | | | |

# PROGRAMMING NOTE:

, C & E

Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.1.2 Inclusion/Exclusion Criteria Enrolled Set

| Subject Number | Date | Inclusion/<br>Exclusion | Criteria Not Met |
|---|---|---|---|
| 12345 | DDMMMXXXX | Inclusion | Inclusion Criteria not met text |
| 12345 | | Exclusion | Exclusion Criteria met text |
| 23456 | DDMMMXXXX | Inclusion | Inclusion Criteria not met text |
| 23456 | | Exclusion | Exclusion Criteria met text |
| 34567 | DDMMMYYYY | Inclusion | Inclusion Criteria not met text |
| 34567 | DDMMMYYYY | Exclusion | Exclusion Criteria met text |

Listing 16.2.1.3 Study Completion Safety Analysis Set

Treatment Sequence: XXX

| | | | Other Reason | Other Reason Specification Text | Other Reason Specification Text | Other Reason Specification Text | |
|---|---|---|---|---|---|---|---|
| | | | Primary Reason for Termination (AE number) Other Reason | Reason Text (AENUM) | Reason Text (AENUM) | Reason Text (AENUM) | |
| Date of | Completion/ | Termination | (Study Day) | ODMIMIYYYY (NN) DDMIMIYYYY (NN) | DDMMMYYYY (NN) | DDMMYYYY (NN) | |
| | Date of Final Completion/ | Contact | (Study Day) | DDMMMYYYY (NN) | DDMMXXXX (NN) | DDMMYYYY (NN) | |
| | | Completed | ber Study | Yes/No | Yes/No | Yes/No | |
| | | | Subject Number Study | 12345 | 23456 | 34567 | : |

# PROGRAMMING NOTE: Exposure unit: days.

Program: XXX.SAS

Listing 16.2.2.1
Protocol Deviations
Enrolled Set


Treatment Sequence: XXX

| Subject Number | Date of Deviation (Study Day) | Classification | Deviation | Deviation Specification |
|---|---|---|---|---|
| 12345<br>23456<br>34567 | DDMMMYYYY (NN)<br>DDMMMYYYY (NN) | Major/Minor<br>Major/Minor<br>Major/Minor | Deviation text Deviation text Deviation text | Deviation specification text Deviation specification text Deviation specification text |

# PROGRAMMING NOTE:

Program: XXX.SAS


Listing 16.2.3.1 Analysis Sets Enrolled Set

Treatment Sequence: XXX

| Subject Number | Enrolled Set | Randomized Set | Safety Analysis Set | PK/PD Analysis Set |
|---|---|---|---|---|
| 12345 | Yes/No | Yes/No | Yes/No | Yes/No |
| 23456 | Yes/No | Yes/No | Yes/No | Yes/No |
| 34567 | Yes/No | Yes/No | Yes/No | Yes/No |
| : | | | | |

# PROGRAMMING NOTE:

Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.4.1 Demographic Data Safety Analysis Set

Treatment Sequence: XXX

| BMI<br>(kg/m2) | N. NN | N.NN | NN.N | |
|---|---|---|---|---|
| Weight<br>(kg) | N. NN | NN.N | N.N | |
| Height (cm) | NN. | NN.N | N.N. | |
| Race | Race | Race | Race | |
| Ethnicity Race | Ethnicity | Ethnicity | Ethnicity | |
| Gender | M/F | M/F | M/F | |
| Age (years)/<br>Date of Birth Gender | NN/<br>DDMMYYYY | NN/<br>DDMMYYYYY | NN/<br>DDMMYYYY | |
| Date/Time of<br>Informed<br>Consent<br>(Study Day) | DDMMMYYYY/<br>HH:MM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) | |
| ICF Version | DDMMYYYY | DDMMMYYYY | DDMMYYYY | |
| Subject<br>Number | 12345 | 23456 | 34567 | : |

# PROGRAMMING NOTE:

Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.4.2 Medical History Safety Analysis Set


Treatment Sequence: XXX

| Start Date<br>Subject Number (Study Day) | Start Date<br>r (Study Day) | End Date<br>(Study Day) /<br>Ongoing? | Body System | System Organ Class /<br>Preferred Term /<br>Verbatim Term |
|---|---|---|---|---|
| 12345 | DDMMYYYY<br>(NN) | DDMMMYYYY<br>(NN) / Ongoing | Body System | System Organ Class<br>/Preferred Term |
| 12345 | DDMMYYYY<br>(NN) | DDMMMYYYY<br>(NN) / Ongoing | Body System | System Organ Class<br>/Preferred Term |
| 23456 | DDMMMYYYY (NN) | DDMMMYYYY<br>(NN) / Ongoing | Body System | System Organ Class<br>/Preferred Term |
| 23456 | DDMMYYYY<br>(NN) | DDMMMYYYY<br>(NN) / Ongoing | Body System | System Organ Class<br>/Preferred Term |
| 34567 | DDMMYYYY<br>(NN) | DDMMMYYYY<br>(NN) / Ongoing | Body System | System Organ Class<br>/Preferred Term |
| 34567 | DDMMMYYYY<br>(NN) | DDMMMYYYY<br>(NN) / Ongoing | Body System | System Organ Class<br>/Preferred Term |
| ÷ | | | | |

# PROGRAMMING NOTE:

Xeris Pharmaceuticals, Inc. DPI-201

Treatment Sequence: XXX

Listing 16.2.4.3
Prior/Concomitant Medications
Safety Analysis Set


| Subject<br>Number | Prior/<br>Concomitant<br>(Treatment<br>Group) | Start Date/<br>Time<br>(Study Day) | End Date/<br>Time<br>(Study Day) /<br>Ongoing? | Medication / Preferred Term / ATC Level 2 / ATC Level 4 | Indication/<br>Reason /<br>Specify | Dose /<br>Unit /<br>Frequency /<br>Route |
|---|---|---|---|---|---|---|
| 12345 | Prior/<br>Concomitant<br>(XXX) | DDMMMYYYY/<br>HH:MM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) / Ongoing | Medication Text<br>/Preferred Term Text<br>/ATC Level 2 Text<br>/ATC Level 4 Text | Reason /<br>Specification Text | Dose<br>/Unit<br>/Frequency<br>/Route |
| 12345 | Prior/<br>Concomitant<br>(XXX) | DDMMMYYYY/<br>HH:MM<br>(NN) | DDWMMYYYY/<br>HH:MM<br>(NN) / Ongoing | Medication Text<br>/Preferred Term Text<br>/ATC Level 2 Text<br>/ATC Level 4 Text | Reason /<br>Specification Text | Dose<br>/Unit<br>/Frequency<br>/Route |
| 23456 | Prior/<br>Concomitant<br>(XXX) | DDMMMYYYY/<br>HH:MM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) / Ongoing | Medication Text<br>/Preferred Term Text<br>/ATC Level 2 Text<br>/ATC Level 4 Text | Reason /<br>Specification Text | Dose<br>/Unit<br>/Frequency<br>/Route |
| 23456 | Prior/<br>Concomitant<br>(XXX) | DDWMMYYYY/<br>HH:MM<br>(NN) | DDWMMYYYY/<br>HH:MM<br>(NN) / Ongoing | Medication Text<br>/Preferred Term Text<br>/ATC Level 2 Text<br>/ATC Level 4 Text | Reason /<br>Specification Text | Dose<br>/Unit<br>/Frequency<br>/Route |
| 34567 | Prior/<br>Concomitant<br>(XXX) | DDMMMYYYY/<br>HH:MM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) / Ongoing | Medication Text<br>/Preferred Term Text<br>/ATC Level 2 Text<br>/ATC Level 4 Text | Reason /<br>Specification Text | Dose<br>/Unit<br>/Frequency<br>/Route |
| 34567 | Prior/<br>Concomitant<br>(XXX) | DDWMYYYY/<br>HH:MM<br>(NN) | DDWMMYYYY/<br>HH:MM<br>(NN) / Ongoing | Medication Text<br>/Preferred Term Text<br>/ATC Level 2 Text<br>/ATC Level 4 Text | Reason /<br>Specification Text | Dose<br>/Unit<br>/Frequency<br>/Route |
| : | | | | | | |

PROGRAMMING NOTE: For 'Other' unit, frequency and route also include text specification.

Xeris Pharmaceuticals, Inc. DPI-201

Treatment Sequence: XXX


Listing 16.2.5.1.1 Exposure Safety Analysis Set

| Subject<br>Number | Visit / Date / Time / (Study Day) | Treatment<br>Administered | Full Dose<br>Administered? | Dose | Reason Dose Adjusted | Dosing Comments |
|---|---|---|---|---|---|---|
| | Visit 1<br>DDWMMYYYY/<br>HH:MM<br>(NN) | XXX | Y/N | NN | Reason Text | Comment text |
| <u> Б П н о</u> | Visit 2<br>DDMMMYYYY/<br>HH:MM<br>(NN) | × | K/N | NN | Reason Text | Comment text |
| | Visit 1<br>DDMMMYYYY/<br>HH:MM<br>(NN) | ×× | Y/N | NN | Reason Text | Comment text |
| | Visit 2<br>DDMMMYYYY/<br>HH:MM<br>(NN) | ××× | ¥/N | NN | Reason Text | Comment text |
| | Visit 1<br>DDMMMYYYY/<br>HH:MM<br>(NN) | × | Y/N | N<br>N | Reason Text | Comment text |
| | Visit 2<br>DDMMMYYYY/<br>HH:MM<br>(NN) | ××× | ¥/N | NN | Reason Text | Comment text |

Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.7.1
Adverse Events
Safety Analysis Set

Treatment Group: XXX

| Subject<br>Number | System Organ Class /<br>Preferred Term /<br>AE Term | TEAE | SAE | Start Date/Time (Study Day) | End Date/Time<br>(Study Day) /<br>Ongoing | Severity | Relation<br>to Study<br>Treatment | Action<br>Taken | Other Ou<br>Action<br>Taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| 12345 | System Organ Class<br>/Preferred Term<br>/Verbatim | K/N | X/N | DDMMXXXY/<br>HH:MM<br>(N) | DDMMMYYYY/<br>HH:MM<br>(N) / Ongoing | Severity | Relation | Action | Y / Specify Outcome | utcome |
| 23456 | System Organ Class<br>/Preferred Term<br>/Verbatim | K/N | X/N | DDMMMYYYY/<br>HH:MM<br>(N) | DDMMMYYYY/<br>HH:MM<br>(N) / Ongoing | Severity | Relation | Action | Y / Specify Outcome | utcome |
| 34567 | System Organ Class<br>/Preferred Term<br>/Verbatim | X/N | N/X | DDMMMYYYY/<br>HH:MM<br>(N) | DDWMMYYYY/<br>HH:WM<br>(N) / Ongoing | Severity | Relation | Action | Y / Specify Outcome | utcome |
| : | | | | | | | | | | |

# PROGRAMMING NOTE:

Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.8.1.1 Vital Sign Data Safety Analysis Set

| XXX |
|-----------------|
| tment Sequence: |
| Treatm |

| Subject<br>Number | Parameter (Unit) | Visit /<br>Timepoint | Treatment<br>Group | Date/Time (Study Day) | Position | Result | Change from<br>Pre-Dose | Clinically<br>Significant | Not Done /<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| 12345 | Parameter 1 (Unit) | Visit 1 /<br>Timepoint X | XXX | DDMMMYYYY/<br>HH:MM<br>(NN) | Position | NN.N | NN.N | No/Yes | |
| 12345 | Parameter 1 (Unit) | Visit 2 /<br>Timepoint X | ××× | DDMMYYYY/<br>HH:MM<br>(NN) | Position | NN.N | NN . N | No/Yes | |
| | Parameter 2 (Unit) | Visit 1 /<br>Timepoint X | XXX | DDMMMYYYY /<br>HH:MM<br>(NN) | Position | NN.N | NN.N | No/Yes | |
| | Parameter 2 (Unit) | Visit 2 /<br>Timepoint X | ××× | DDMMYYYY/<br>HH:MM<br>(NN) | Position | NN.N | NN.N | No/Yes | |
| | Parameter 3 (Unit) | Visit 1 /<br>Timepoint X | XXX | DDMMMYYYY/<br>HH:MM<br>(NN) | Position | NN.N | NN.N | No/Yes | |
| | Parameter 3 (Unit) | Visit 2 /<br>Timepoint X | ××× | DDMMYYYY/<br>HH:MM<br>(NN) | Position | NN.N | N. NN | No/Yes | |
| | Parameter 4 (Unit) | Visit 1 /<br>Timepoint X | XXX | DDMMMYYYY/<br>HH:MM<br>(NN) | Position | NN.N | NN.N | No/Yes | |
| | Parameter 4 (Unit) | Visit 2 /<br>Timepoint X | XXX | DDMMYYYY/<br>HH:MM<br>(NN) | Position | NN. | NN.NN | No/Yes | |
| : | | | | | | | | | |

Listing 16.2.8.2.1 Physical Examination Data Safety Analysis Set Confidential

Treatment Sequence: XXX

| Subject<br>Number | Parameter (Unit) | Visit | Treatment<br>Group | Date/Time (Study Day) | Result | Reason |
|---|---|---|---|---|---|---|
| 12345 | Parameter 1 | Visit 1 | × | DDMMYYYY/<br>HH:MM<br>(NN) | Normal /<br>Abnormal NCS /<br>Abnormal CS /<br>Not Done | |
| | Parameter 2 | Visit 1 | XXX | DDMMYYYY/<br>HH:MM<br>(NN) | Normal /<br>Abnormal NCS /<br>Abnormal CS /<br>Not Done | |
| | Parameter 3 | Visit 1 | XXX | DDMMYYYY/<br>HH:MM<br>(NN) | Normal /<br>Abnormal NCS /<br>Abnormal CS /<br>Not Done | |
| | Parameter 4 | Visit 1 | × | DDMMYYYYY/<br>HH:MM<br>(NN) | Normal /<br>Abnormal NCS /<br>Abnormal CS /<br>Not Done | |
| : | | | | | | |

Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.8.3.1 Hematology Data Safety Analysis Set

Treatment Sequence: XXX

| Subject<br>Number | Parameter (Unit) | Visit | Date/Time (Study Day) | Result | Normal Range | Reference Range<br>Indicator | Change from Not Done /<br>Baseline Reason |
|---|---|---|---|---|---|---|---|
| 12345 | Parameter 1 (Unit) | Visit 1 | DDMMYYYY<br>HH:MM<br>(NN) | NN.N | LL.L - HH.H | Low/Normal/High | NN . N |
| 12345 | Parameter 1 (Unit) | Visit 2 | DDMMYYYY<br>HH:MM<br>(NN) | NN.N | тг.т - нн.н | Low/Normal/High | NN . N |
| | Parameter 2 (Unit) | Visit 1 | DDMMYYYY<br>HH:MM<br>(NN) | NN.N | LL.L - НН.Н | Low/Normal/High | NN. N |
| | Parameter 2 (Unit) | Visit 2 | DDMMYYYY<br>HH:MM<br>(NN) | NN.N | л.т - нн.н | Low/Normal/High | NN . N |
| | Parameter 3 (Unit) | Visit 1 | DDMMYYYY<br>HH:MM<br>(NN) | NN.N | LL.L - НН.Н | Low/Normal/High | NN.N |
| | Parameter 3 (Unit) | Visit 2 | DDMMYYYY<br>HH:MM<br>(NN) | NN.N | л.т - нн.н | Low/Normal/High | NN . N |
| | Parameter 4 (Unit) | Visit 1 | DDMMYYYY<br>HH:MM<br>(NN) | NN.N | LL.L - НН.Н | Low/Normal/High | NN. N |
| : | Parameter 4 (Unit) | Visit 2 | DDMMYYYY<br>HH:MM<br>(NN) | Z. | тг.г - нн.н | Low/Normal/High | NN . N |

Page X of Y Confidential Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.8.3.2 Serum Chemistry Data Safety Analysis Set

PROGRAMMING NOTE: Same shell as Listing 16.2.8.3.1.

Treatment Sequence: XXX

Worldwide Clinical Trials DDMMMYYYY:HH:MM Program: XXX.SAS Page X of Y Confidential Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.8.3.3 C-Peptide and HbAlc Data Safety Analysis Set

PROGRAMMING NOTE: Same shell as Listing 16.2.8.3.1.

Treatment Sequence: XXX

Worldwide Clinical Trials DDMMMYYYY:HH:MM Program: XXX.SAS

Xeris Pharmaceuticals, Inc. DPI-201

Treatment Sequence: XXX


Listing 16.2.8.3.4 Urine Drug Screen Data Safety Analysis Set

| Subject Number | Parameter (Unit) | Visit | Date (Study Day) | Result | Not Done /<br>Reason |
|---|---|---|---|---|---|
| 12345 | Parameter 1 (Unit) | Visit 1 | DDMMMYYYY<br>HH:MM | XXX | |
| 12345 | Parameter 1 (Unit) | Visit 2 | (NN)<br>DDMMYYYY<br>HH:MM<br>(NN) | XXX | |
| | Parameter 2 (Unit) | Visit 1 | DDMMYYYY<br>HH:MM | XXX | |
| | Parameter 2 (Unit) | Visit 2 | (NN)<br>DDMMAYYYY<br>HH:MM<br>(NN) | ××× | |
| | Parameter 3 (Unit) | Visit 1 | DDMMYYYYY<br>HH:MM<br>(NN) | ×× | |
| | Parameter 3 (Unit) | Visit 2 | DDMMYYYY<br>HH:MM<br>(NN) | XXX | |
| | Parameter 4 (Unit) | Visit 1 | DDMMYYYY<br>HH: MM | XXX | |
| | Parameter 4 (Unit) | Visit 2 | (NN)<br>DDWMYYYY<br>HH:MM<br>(NN) | ××× | |
| ÷ | | | | | |

Page X of Y Confidential Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.8.3.5 Urine Pregnancy Test Data Safety Analysis Set

PROGRAMMING NOTE: Same shell as Listing 16.2.8.3.4.

Treatment Sequence: XXX

Worldwide Clinical Trials DDMMMYYYY:HH:MM Program: XXX.SAS

Xeris Pharmaceuticals, Inc. DPI-201

Treatment Sequence: XXX


Listing 16.2.8.4.1 ECG Data Safety Analysis Set

| Subject<br>Number | Parameter (Unit) | Visit | Date/Time (Study Day) | Position | Result | Not Done /<br>Reason |
|---|---|---|---|---|---|---|
| 12345 | Parameter 1 (Unit) | Visit 1 | DDMMYYYY/<br>HH: MM<br>(NN) | Position | NN.N / Normal / Abnormal (NCS) / Abnormal (CS) | |
| 12345 | Parameter 1 (Unit) | Visit 2 | DDMMMYYYY /<br>HH: MM<br>(NN) | Position | | |
| | Parameter 2 (Unit) | Visit 1 | DDMMYYYYY/<br>HH:MM<br>(NN) | Position | NN.N / Normal / Abnormal (NCS) / Abnormal (CS) | |
| | Parameter 2 (Unit) | Visit 2 | DDMMMYYYY/<br>HH:MM<br>(NN) | Position | | |
| | Parameter 3 (Unit) | Visit 1 | DDMMYYYY/<br>HH:MM<br>(NN) | Position | NN.N / Normal / Abnormal (NCS) / Abnormal (CS) | |
| | Parameter 3 (Unit) | Visit 2 | DDMMYYYY/<br>HH: MM<br>(NN) | Position | | |
| : | | | | | | |

PROGRAMMING NOTE: For overall interpretation add also ECG Interpretation Text together with the result.

Program: XXX.SAS

Safety Analysis Set Listing 16.2.8.5.1 Draize Scale Data

Treatment Sequence: XXX

PROGRAMMING NOTE: Same shell as Listing 16.2.8.2.1 but without 'Clinically Significant' and 'Not Done' columns.

PROGRAMMING NOTE: Results are as follows for Erythema Formation:

0 - No erythema

1 - Very slight erythema2 - Well defined erythema

3 - Moderate erythema

4 - Severe erythema

and for Edema Formation:

0 - No edema

Very slight edema
 Slight edema
 Moderate edema
 Severe edema

Page X of

Listing 16.2.8.6.1 Injection Site Discomfort Assessment Data Safety Analysis Set

Treatment Sequence: XXX

PROGRAMMING NOTE: Same shell as Listing 16.2.8.2.1 but without 'Clinically Significant' column.

PROGRAMMING NOTE: Add possible comment together with result.

PROGRAMMING NOTE: Results include:

11 point numeric rating scale.

1a. How would you describe any discomfort you felt from the study drug? (Check all that apply):

None (Please ignore question 1b.)

Pain (eg, throbbing, soreness, muscle ache)

Itching

Tingling, twitching, or numbness

Irritation (eg, burning, stinging)

Other

1b. About how long did the discomfort last after the injection? (Check one):

Less than 1 minute

1-2 minutes

3-5 minutes

5-5 minutes 6-9 minutes at least 10 minutes (Please complete question 1c before leaving the clinic.)

1c. In total, how long did the discomfort last after the injection? (Please enter a number below):

Minutes


Listing 16.2.8.7.1
Plasma Glucose Concentration Data Safety Analysis Set

Treatment Sequence: XXX

Xeris Pharmaceuticals, Inc. DPI-201

| amplect Namber | VISIC | Treatment Group | Date (Study Day) | T.me | Kesult<br>( <unit>)</unit> | Not Done /<br>Reason |
|---|---|---|---|---|---|---|
| 12345 | Visit 1 | XXX | DDMMXXXX (NN) | HH: MM | N. NN | |
| | | | | HH: MM | N. NN | |
| | | | | HH: MM | N.NN | |
| | | | | HH: MM | N. NN | |
| | | | | HH:MM | NN.N | |

PROGRAMMING NOTE: Visits: 'Visit 2', 'Visit 3', 'Visit 4'.

Xeris Pharmaceuticals, Inc. DPI-201

Listing 16.2.8.7.2
Plasma Glucose PD Parameter Data Safety Analysis Set

Treatment Sequence: XXX

| Subject Number | Visit | Treatment Group | Parameter | Result | Not Done /<br>Reason |
|---|---|---|---|---|---|
| 12345 | Visit 1 | XXX | Parameter 1 (Unit) | N.NN | |
| 12345 | Visit 1 | XXX | Parameter 2 (Unit) | NN.NN | |
| 12345 | Visit 1 | XXX | Parameter 3 (Unit) | NN.N | |
| 12345 | Visit 1 | XXX | Parameter 4 (Unit) | N.NN | |
| 12345 | Visit 1 | XXX | Parameter 5 (Unit) | N.NN | |
| 12345 | Visit 1 | XXX | Parameter 6 (Unit) | N.NN | |
| 12345 | Visit 1 | XXX | Parameter 7 (Unit) | NN.N | |
| 12345 | Visit 1 | XXX | Parameter 8 (Unit) | N.NN | |
| : | | | | | |

PROGRAMMING NOTE: Include parameters as specified in the Statistical Analysis Plan.

Xeris Pharmaceuticals, Inc. DPI-201

Treatment Sequence: XXX


Listing 16.2.8.7.3 Glucose Challenge Safety Analysis Set

| Subject Number Visit | Visit | Treatment Group | Date/Time (Study Day) Date/Time (Study Day) of Challenge Start of Challenge End | Date/Time (Study Day)<br>of Challenge End | Did subject complete<br>100% of Glucose<br>Challenge | Amount of Glucose<br>Challenge Complete (%) |
|---|---|---|---|---|---|---|
| 12345 | Visit 1 | XXX | DDMMMYYYY/<br>HH:NM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) | No/Yes | NN |
| 12345 | Visit 2 | XXX | DDMMYYYY/<br>HH:MM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) | No/Yes | NN |
| 12345 | Visit 3 | XXX | DDMMMYYYY/<br>HH:MM<br>(NN) | DDMMMYYYY/<br>HH:MM<br>(NN) | No/Yes | NM |
| : | | | | | | |

# PROGRAMMING NOTE:

Confidential Xeris Pharmaceuticals, Inc. DPI-201

Page X of Y

Listing 16.2.8.8.1 Hypoglycemic Events Safety Analysis Set

Treatment Sequence: XXX

| | Ĵξ | 7 | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Time to Resolution of | Hypo Event after IV | Dextrose<br>Administration | (minutes) | NN | NN | NN | |
| Time to IV Dextrose | Administration | (minutes) | (Amount of IV Dextrose (g) needed for BG>70 | mg/dL) | NN * NN | NN × NN | NN × NN | |
| | | | Time to Hypo Event | (minutes) | *NN | *NN | * NN | |
| | | | | Treatment Group Experienced Hypo Event | No/Yes | No/Yes | No/Yes | |
| | | | | Treatment Group | XXX | XXX | XXX | |
| | | | | oer Visit | Visit 1 | Visit 2 | Visit 3 | |
| | | | | Subject Number Visit | 12345 | 12345 | 12345 | : |

### PROGRAMMING NOTE:

If hypo event occurs after glucose challenge then it will not be included as event and will be censored at the time of glucose challenge. Only events occurring after treatment and prior to glucose challenge are included as events.


 $Figure \ 14.3.1.1 \\ Time \ (\mbox{minutes}) \ \mbox{to IV Dextrose Administration from Study Drug Administration by Treatment Group \\$ Safety Analysis Set



Figure 14.3.1.2 Time (minutes) to Hypoglycemic Event from Study Drug Administration by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Figure 14.3.1.1.

Figure 14.3.1.3 Time (minutes) to Resolution of Hypoglycemic Event from IV Dextrose Administration by Treatment Group Safety Analysis Set

PROGRAMMING NOTE: Same shell as Figure 14.3.1.1.


Figure 14.5.1.1
Plasma Glucose Concentration Data, Mean Profiles on Linear Scale
PD Analysis Set



# PROGRAMMING NOTE:

Xeris Pharmaceuticals, Inc. DPI-201

Figure 14.5.1.2 Plasma Glucose Concentration Data, Individual Profiles on Linear Scale PD Analysis Set

Treatment: XXX



PROGRAMMING NOTE: Repeat for treatments 'XP-3924', 'Regular Insulin', 'Regular Insulin + Pramlintide'.

Program: XXX.SAS



#### **Certificate Of Completion**

Envelope Id: BC295336D9504C59B86A748098257AEB

Subject: Please DocuSign: DPI-201 SAP v1.0 2019-11-14 sponsor signed.pdf

Source Envelope:

Document Pages: 116Signatures: 2Envelope Originator:Certificate Pages: 2Initials: 0Tuomas KemppainenAutoNav: Enabled3800 Paramount Parkway

Envelopeld Stamping: Disabled

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Suite 400

Status: Completed

Morrisville, NC 27560

tuomas.kemppainen@worldwide.com

IP Address: 91.152.17.218

Sent: 15-Nov-2019 | 08:58

Viewed: 15-Nov-2019 | 09:30

Signed: 15-Nov-2019 | 13:58

Sent: 15-Nov-2019 | 08:58

Viewed: 15-Nov-2019 | 09:14

Signed: 15-Nov-2019 | 09:21

#### **Record Tracking**

Status: Original

15-Nov-2019 | 08:56

Holder: Tuomas Kemppainen

tuomas.kemppainen@worldwide.com

Location: DocuSign

**Timestamp** 

#### Signer Events

Ioulietta Mulligan

ioulietta.mulligan@worldwide.com

Manager Biostatistics Worldwide Clinical Trials

Security Level: Email, Account Authentication

(Required)

Signature

Ioulietta Mulligan

·

Signature Adoption: Pre-selected Style

Signature ID:

E2F77940-2D67-46B3-BD21-46FE31684871

Using IP Address: 86.132.133.142

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I have reviewed this document

#### Electronic Record and Signature Disclosure:

Not Offered via DocuSign

Tuomas Kemppainen

tuomas.kemppainen@worldwide.com

Senior Statistical Programmer Worldwide Clinical Trials

Security Level: Email, Account Authentication

(Required)

Tunken

Signature Adoption: Uploaded Signature Image

Signature ID:

1555D305-747C-4F48-8CA5-46AD81C72A6E

Using IP Address: 91.152.17.218

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I have reviewed this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

In Person Signer Events

Signature Timestamp

Editor Delivery Events Status Timestamp

Agent Delivery Events Status Timestamp

Intermediary Delivery Events Status Timestamp

Certified Delivery Events Status Timestamp

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 15-Nov-2019 08:58 |
| Certified Delivered | Security Checked | 15-Nov-2019 09:30 |
| Signing Complete | Security Checked | 15-Nov-2019 13:58 |
| Signing Complete Completed | Security Checked<br>Security Checked | 15-Nov-2019 13:58<br>15-Nov-2019 13:58 |